CLINICAL TRIAL: NCT02251704
Title: An Epidemiology Study to Assess Plasmodium Falciparum Parasite Prevalence and Malaria Control Measures in Catchment Areas of Two Interventional Studies Pre- and Post RTS,S/AS01E Introduction (EPI MAL-002 and EPI-MAL-003) to Assess, in Field Conditions, Vaccine Benefit: Risk in Children in Sub Saharan Africa
Brief Title: Epidemiology Study of Malaria Transmission Intensity in Sub-Saharan Africa
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: The PATH Malaria Vaccine Initiative (MVI) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 116682
Record Dates: First submitted 2014-09-25; First posted 2014-09-29 (Estimated); Results first posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Malaria; Malaria Vaccines
Keywords: Malaria; MTI; Surveillance study; Africa; RTS,S/AS01; Epidemiology; Plasmodium falciparum; Malaria control interventions
MeSH Terms: conditions — Malaria; Malaria, Falciparum | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (10):
- Survey 1 Group (Other): Participants aged 6 months to <10 years, enrolled in the current EPI-MAL-005 study from sites that participated in EPI-MAL-002/-003, during study Year 1.
  Interventions: Diagnostic Test: Assessment of body temperature; Procedure: Blood sampling
- Survey 2 Group (Other): Participants aged 6 months to <10 years, enrolled in the current EPI-MAL-005 study from sites that participated in EPI-MAL-002/-003, during study Year 2.
  Interventions: Diagnostic Test: Assessment of body temperature; Procedure: Blood sampling
- Survey 3 Group (Other): Participants aged 6 months to <10 years, enrolled in the current EPI-MAL-005 study from sites that participated in EPI-MAL-002/-003, during study Year 3.
  Interventions: Diagnostic Test: Assessment of body temperature; Procedure: Blood sampling
- Survey 4 Group (Other): Participants aged 6 months to <10 years, enrolled in the current EPI-MAL-005 study from sites that participated in EPI-MAL-002/-003, during study Year 4.
  Interventions: Diagnostic Test: Assessment of body temperature; Procedure: Blood sampling
- Survey 5 Group (Other): Participants aged 6 months to <10 years, enrolled in the current EPI-MAL-005 study from sites that participated in EPI-MAL-002/-003, during study Year 5.
  Interventions: Diagnostic Test: Assessment of body temperature; Procedure: Blood sampling
- Survey 6 Group (Other): Participants aged 6 months to <10 years, enrolled in the current EPI-MAL-005 study from sites that participated in EPI-MAL-002/-003, during study Year 6.
  Interventions: Diagnostic Test: Assessment of body temperature; Procedure: Blood sampling
- Survey 7 Group (Other): Participants aged 6 months to <10 years, enrolled in the current EPI-MAL-005 study from sites that participated in EPI-MAL-002/-003, during study Year 7.
  Interventions: Diagnostic Test: Assessment of body temperature; Procedure: Blood sampling
- Survey 8 Group (Other): Participants aged 6 months to <10 years, enrolled in the current EPI-MAL-005 study from sites that participated in EPI-MAL-002/-003, during study Year 8.
  Interventions: Diagnostic Test: Assessment of body temperature; Procedure: Blood sampling
- Survey 9 Group (Other): Participants aged 6 months to <10 years, enrolled in the current EPI-MAL-005 study from sites that participated in EPI-MAL-002/-003, during study Year 9.
  Interventions: Diagnostic Test: Assessment of body temperature; Procedure: Blood sampling
- Survey 10 Group (Other): Participants aged 6 months to <10 years, enrolled in the current EPI-MAL-005 study from sites that participated in EPI-MAL-002/-003, during study Year 10.
  Interventions: Diagnostic Test: Assessment of body temperature; Procedure: Blood sampling

INTERVENTIONS:
Diagnostic Test: Assessment of body temperature — Axillary body temperature of all participants recorded by a digital thermometer at the time of survey.
Procedure: Blood sampling — Capillary blood samples collected by finger/heel prick for determination of parasite prevalence at the time of survey.

SUMMARY:
This epidemiology study was conducted in parallel with the EPI-MAL-002 (NCT02374450) and EPI-MAL-003 (NCT03855995) studies, enrolling participants from the same health and demographic surveillance system (HDSS) (or equivalent system) populations. The co-primary objectives were to produce longitudinal estimates of parasite prevalence in humans and to record the usage of malaria control measures in areas where the EPI-MAL-002 and EPI-MAL-003 studies were conducted.

DETAILED DESCRIPTION:
This study involved 10 annual cross-sectional surveys conducted during malaria peak transmission seasons. The surveys provided point estimates of parasite prevalence and subsequently enabled a longitudinal assessment of the level of endemicity in each area covered by EPI-MAL-002 and EPI-MAL-003. The study was conducted in parallel with EPI-MAL-002 and EPI-MAL-003 to assess parasite prevalence and malaria control measures before (EPI-MAL-002) and after (EPI-MAL-003) vaccine introduction.

By taking into account variations in malaria transmission intensity (MTI) and malaria control intervention coverage, it enabled a more complete assessment of the benefits and risks of the vaccine introduction, and thereby provided greater insight into the potential vaccine impact in EPI-MAL-002/-003 by adjusting incidence data for overall changes in transmission and other malaria control intervention coverage, and assisted in the generalisation of results to other populations.

ELIGIBILITY:
Inclusion Criteria:

* Participants whose parent(s)/Legally Acceptable Representative(s) [LAR(s)], in the opinion of the investigator, could and would comply with the requirements of the protocol.
* A male or female aged 6 months to under 10 years at the time of the survey.
* Signed informed consent or thumb-printed and witnessed informed consent was obtained from the parent(s)/LAR(s) of the child.

Exclusion Criteria:

* Child was in care.
* Had current active participation in any trial involving administration of an investigational malaria vaccine or malaria drug.

Ages: 6 Months to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54115 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2024-07-06 (Actual); Study Completion 2024-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- Burkina Faso (2):
  - GSK Investigational Site, Nouna
  - GSK Investigational Site, Ouagadougou
- Ghana (2):
  - GSK Investigational Site, Kintampo
  - GSK Investigational Site, Navrongo
- Kenya (2):
  - GSK Investigational Site, Kisumu
  - GSK Investigational Site, Nairobi
- Malawi (2):
  - GSK Investigational Site, Chikwawa
  - GSK Investigational Site, Mangochi
- GSK Investigational Site, Dakar, Senegal
- GSK Investigational Site, Amani, Tanzania

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from Health and Demographic Surveillance System (HDSS) (or equivalent system) catchment areas at the sites participating in the EPI-MAL-002 (NCT02374450) and EPI-MAL-003 (NCT03855995) studies of the candidate malaria vaccine RTS,S/AS01E in sub-Saharan Africa.
Pre-assignment Details: Out of 54115 participants enrolled, 54100 participants were included in the Total Effective Cohort and started the study.
Period: Overall Study
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group
Started | 4214 | 4204 | 2400 | 3003 | 5417 | 5991 | 7246 | 7220 | 7203 | 7202
Completed | 4214 | 4204 | 2400 | 3003 | 5417 | 5991 | 7246 | 7220 | 7203 | 7202
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline analysis was performed on the Total Effective Cohort, which included all participants enrolled in the study for whom data was collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group | Total
Number analyzed (Participants) | 4214 | 4204 | 2400 | 3003 | 5417 | 5991 | 7246 | 7220 | 7203 | 7202 | 54100
Age, Continuous [Mean (Standard Deviation); unit: Years] — The Age Continuous analysis was based on participants' age recorded at the time of signing the Informed Consent Form (ICF). Population: The Age Continuous analysis is presented separately for each of the 10-survey year.
  Years
    Year 1: number analyzed (Participants) | 4214 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4214
    Year 1 | 4.0 (2.8) |  |  |  |  |  |  |  |  |  | 4.0 (2.8)
    Year 2: number analyzed (Participants) | 0 | 4204 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4204
    Year 2 |  | 4.0 (2.7) |  |  |  |  |  |  |  |  | 4.0 (2.7)
    Year 3: number analyzed (Participants) | 0 | 0 | 2400 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2400
    Year 3 |  |  | 4.0 (2.8) |  |  |  |  |  |  |  | 4.0 (2.8)
    Year 4: number analyzed (Participants) | 0 | 0 | 0 | 3003 | 0 | 0 | 0 | 0 | 0 | 0 | 3003
    Year 4 |  |  |  | 4.0 (2.8) |  |  |  |  |  |  | 4.0 (2.8)
    Year 5: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5417 | 0 | 0 | 0 | 0 | 0 | 5417
    Year 5 |  |  |  |  | 4.1 (2.7) |  |  |  |  |  | 4.1 (2.7)
    Year 6: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 5991 | 0 | 0 | 0 | 0 | 5991
    Year 6 |  |  |  |  |  | 4.0 (2.7) |  |  |  |  | 4.0 (2.7)
    Year 7: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7246 | 0 | 0 | 0 | 7246
    Year 7 |  |  |  |  |  |  | 4.1 (2.7) |  |  |  | 4.1 (2.7)
    Year 8: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7220 | 0 | 0 | 7220
    Year 8 |  |  |  |  |  |  |  | 4.0 (2.7) |  |  | 4.0 (2.7)
    Year 9: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7203 | 0 | 7203
    Year 9 |  |  |  |  |  |  |  |  | 4.0 (2.7) |  | 4.0 (2.7)
    Year 10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7202 | 7202
    Year 10 |  |  |  |  |  |  |  |  |  | 4.0 (2.7) | 4.0 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2053 | 2090 | 1191 | 1448 | 2642 | 2963 | 3626 | 3660 | 3505 | 3593 | 26771
  Male | 2161 | 2114 | 1209 | 1555 | 2775 | 3028 | 3620 | 3560 | 3698 | 3609 | 27329
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Infected With Plasmodium Falciparum (P. Falciparum) by World Health Organisation (WHO) Age Group
Description: The number of participants was summarized by the WHO age group (0.5-1 year [Y] and 2-9Y) and by center number/ country [Burkina Faso (BF), Senegal (SN), Tanzania (TZ), Kenya (KE), Ghana (GH), Malawi (MA)]/ city. Unexposed (UNEXP) sites are the ones in which the RTS,S vaccine was not planned to be implemented during the course of the study however, vaccinated participants could still have been randomly selected in this population if vaccination happened in an exposed (EXP) site, due to cross-site migration. The infection was identified using a blood smear slide and determined using microscopy.
Time Frame: At Day 1 (survey completion visit)
Population: The analysis was performed on the According To Protocol (ATP) Cohort which included all participants who met the eligibility criteria, adhered to the procedures defined in the protocol, had no elimination criteria during the study, had at least one laboratory result from a blood sample available and with usable data for the specified analysis at the specified time point. Here, 'number analyzed' = participants with available data for each specified row.
Measure: Count of Participants; unit: Participants
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group
Number analyzed (Participants) | 424 | 425 | 420 | 430 | 431 | 430 | 442 | 427 | 427 | 427
Participants
  0.5-1Y, 207078_BF_Nouna: number analyzed (Participants) | 182 | 186 | 180 | 182 | 0 | 0 | 0 | 0 | 0 | 0
  0.5-1Y, 207078_BF_Nouna | 98 | 148 | 82 | 46 |  |  |  |  |  |
  0.5-1Y, 207079_BF_Sapone: number analyzed (Participants) | 182 | 176 | 182 | 178 | 0 | 0 | 0 | 0 | 0 | 0
  0.5-1Y, 207079_BF_Sapone | 46 | 54 | 22 | 31 |  |  |  |  |  |
  0.5-1Y, 207080_SN_Niakhar: number analyzed (Participants) | 186 | 176 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  0.5-1Y, 207080_SN_Niakhar | 2 | 0 |  |  |  |  |  |  |  |
  0.5-1Y, 207081_TZ_Korogwe: number analyzed (Participants) | 184 | 178 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  0.5-1Y, 207081_TZ_Korogwe | 6 | 2 |  |  |  |  |  |  |  |
  0.5-1Y, 207082_KE_Kombewa: number analyzed (Participants) | 183 | 181 | 182 | 182 | 183 | 180 | 180 | 183 | 181 | 181
  0.5-1Y, 207082_KE_Kombewa | 32 | 47 | 47 | 46 | 44 | 47 | 27 | 26 | 27 | 17
  0.5-1Y, 207083_GH_Kintampo: number analyzed (Participants) | 180 | 181 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  0.5-1Y, 207083_GH_Kintampo | 33 | 36 |  |  |  |  |  |  |  |
  0 .5-1Y, 207083_GH_Kintampo_EXP: number analyzed (Participants) | 0 | 0 | 182 | 182 | 180 | 180 | 180 | 178 | 176 | 181
  0 .5-1Y, 207083_GH_Kintampo_EXP |  |  | 41 | 42 | 22 | 20 | 14 | 10 | 6 | 3
  0.5-1Y, 207083_GH_Kintampo_UNEXP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 180 | 178 | 181 | 180 | 181
  0.5-1Y, 207083_GH_Kintampo_UNEXP |  |  |  |  |  | 29 | 22 | 15 | 17 | 8
  0.5-1Y, 207084_SN_Keur Soce: number analyzed (Participants) | 181 | 176 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  0.5-1Y, 207084_SN_Keur Soce | 0 | 1 |  |  |  |  |  |  |  |
  0 .5-1Y, 228607_GH_Navrongo_EXP: number analyzed (Participants) | 0 | 0 | 0 | 170 | 178 | 181 | 179 | 182 | 177 | 182
  0 .5-1Y, 228607_GH_Navrongo_EXP |  |  |  | 7 | 7 | 7 | 3 | 4 | 8 | 4
  0.5-1Y, 228607_GH_Navrongo_UNEXP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 181 | 177 | 181 | 180 | 186
  0.5-1Y, 228607_GH_Navrongo_UNEXP |  |  |  |  |  | 9 | 9 | 5 | 7 | 4
  0 .5-1Y, 233149_MA_Mangochi: number analyzed (Participants) | 0 | 0 | 0 | 0 | 172 | 173 | 172 | 173 | 174 | 177
  0 .5-1Y, 233149_MA_Mangochi |  |  |  |  | 16 | 7 | 9 | 15 | 4 | 3
  0 .5-1Y, 233150_MA_Chikwawa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 160 | 0 | 179 | 175 | 182 | 180
  0 .5-1Y, 233150_MA_Chikwawa |  |  |  |  | 7 | 0 | 12 | 2 | 1 | 3
  0 .5-1Y, 233149_MA_Monkey Bay: number analyzed (Participants) | 0 | 0 | 0 | 0 | 175 | 172 | 171 | 181 | 178 | 172
  0 .5-1Y, 233149_MA_Monkey Bay |  |  |  |  | 11 | 1 | 6 | 6 | 5 | 8
  0 .5-1Y, 233150_MA_St Monfort: number analyzed (Participants) | 0 | 0 | 0 | 0 | 162 | 0 | 182 | 185 | 180 | 183
  0 .5-1Y, 233150_MA_St Monfort |  |  |  |  | 3 |  | 9 | 1 | 0 | 2
  0 .5-1Y, 235578_KE_Bondo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 180 | 168 | 181 | 180 | 181 | 180
  0 .5-1Y, 235578_KE_Bondo |  |  |  |  | 28 | 32 | 29 | 15 | 19 | 13
  0 .5-1Y, 235578_KE_Gem: number analyzed (Participants) | 0 | 0 | 0 | 0 | 183 | 172 | 180 | 181 | 178 | 181
  0 .5-1Y, 235578_KE_Gem |  |  |  |  | 31 | 20 | 13 | 20 | 20 | 13
  0.5-1Y, 235579_KE_Nyando: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 175 | 176 | 180 | 183 | 181
  0.5-1Y, 235579_KE_Nyando |  |  |  |  |  | 32 | 18 | 15 | 15 | 13
  2-9Y, 207078_BF_Nouna: number analyzed (Participants) | 424 | 414 | 420 | 418 | 0 | 0 | 0 | 0 | 0 | 0
  2-9Y, 207078_BF_Nouna | 305 | 340 | 270 | 211 |  |  |  |  |  |
  2-9Y, 207079_BF_Sapone: number analyzed (Participants) | 422 | 423 | 418 | 422 | 0 | 0 | 0 | 0 | 0 | 0
  2-9Y, 207079_BF_Sapone | 253 | 262 | 172 | 173 |  |  |  |  |  |
  2-9Y, 207080_SN_Niakhar: number analyzed (Participants) | 412 | 425 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  2-9Y, 207080_SN_Niakhar | 7 | 3 |  |  |  |  |  |  |  |
  2-9Y, 207081_TZ_Korogwe: number analyzed (Participants) | 417 | 422 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  2-9Y, 207081_TZ_Korogwe | 57 | 16 |  |  |  |  |  |  |  |
  2-9Y, 207082_KE_Kombewa: number analyzed (Participants) | 416 | 418 | 417 | 418 | 417 | 420 | 420 | 417 | 419 | 419
  2-9Y, 207082_KE_Kombewa | 164 | 142 | 166 | 165 | 143 | 138 | 107 | 97 | 97 | 101
  2-9Y, 207083_GH_Kintampo: number analyzed (Participants) | 420 | 419 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  2-9Y, 207083_GH_Kintampo | 181 | 176 |  |  |  |  |  |  |  |
  2-9Y, 207083_GH_Kintampo_EXP: number analyzed (Participants) | 0 | 0 | 418 | 418 | 420 | 420 | 420 | 422 | 424 | 419
  2-9Y, 207083_GH_Kintampo_EXP |  |  | 184 | 144 | 131 | 99 | 89 | 64 | 57 | 49
  2-9Y, 207083_GH_Kintampo_UNEXP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 420 | 422 | 419 | 420 | 419
  2-9Y, 207083_GH_Kintampo_UNEXP |  |  |  |  |  | 126 | 111 | 84 | 74 | 59
  2-9Y, 207084_SN_Keur Soce: number analyzed (Participants) | 419 | 424 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  2-9Y, 207084_SN_Keur Soce | 3 | 5 |  |  |  |  |  |  |  |
  2-9Y, 228607_GH_Navrongo_EXP: number analyzed (Participants) | 0 | 0 | 0 | 430 | 427 | 418 | 421 | 417 | 423 | 418
  2-9Y, 228607_GH_Navrongo_EXP |  |  |  | 93 | 103 | 90 | 74 | 65 | 66 | 70
  2-9Y, 228607_GH_Navrongo_UNEXP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 419 | 423 | 419 | 420 | 414
  2-9Y, 228607_GH_Navrongo_UNEXP |  |  |  |  |  | 97 | 86 | 70 | 82 | 91
  2-9Y, 233149_MA_Mangochi: number analyzed (Participants) | 0 | 0 | 0 | 0 | 425 | 429 | 427 | 427 | 427 | 424
  2-9Y, 233149_MA_Mangochi |  |  |  |  | 82 | 79 | 42 | 63 | 39 | 61
  2-9Y, 233149_MA_Monkey Bay: number analyzed (Participants) | 0 | 0 | 0 | 0 | 423 | 428 | 429 | 419 | 421 | 427
  2-9Y, 233149_MA_Monkey Bay |  |  |  |  | 52 | 34 | 28 | 32 | 39 | 40
  2-9Y, 233150_MA_Chikwawa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 423 | 0 | 442 | 425 | 418 | 417
  2-9Y, 233150_MA_Chikwawa |  |  |  |  | 62 |  | 85 | 30 | 16 | 22
  2-9Y, 233150_MA_St Monfort: number analyzed (Participants) | 0 | 0 | 0 | 0 | 422 | 0 | 431 | 415 | 420 | 420
  2-9Y, 233150_MA_St Monfort |  |  |  |  | 35 |  | 44 | 13 | 2 | 2
  2-9Y, 235578_KE_Bondo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 431 | 430 | 423 | 426 | 422 | 420
  2-9Y, 235578_KE_Bondo |  |  |  |  | 130 | 147 | 110 | 112 | 86 | 73
  2-9Y, 235578_KE_Gem: number analyzed (Participants) | 0 | 0 | 0 | 0 | 416 | 416 | 424 | 425 | 422 | 421
  2-9Y, 235578_KE_Gem |  |  |  |  | 115 | 111 | 102 | 86 | 90 | 75
  2-9Y, 235579_KE_Nyando: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 425 | 424 | 426 | 417 | 419
  2-9Y, 235579_KE_Nyando |  |  |  |  |  | 121 | 89 | 59 | 79 | 76

2. Secondary Outcome: Number of Participants Infected With P. Falciparum by Center, Gender and Infection Status
Description: The number of participants was summarized by: center number/ country [BF, SN, TZ, KE, GH, MA]/ city, gender (female, male) and infection status (infected, not infected).
Time Frame: At Day 1 (survey completion visit)
Population: The analysis was performed on the ATP Cohort which included all participants who met the eligibility criteria, adhered to the procedures defined in the protocol, had no elimination criteria during the study, had at least one laboratory result from a blood sample available and with usable data for the specified analysis at the specified time point. Here, 'number analyzed' = participants with available data for each specified row.
Measure: Count of Participants; unit: Participants
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group
Number analyzed (Participants) | 606 | 601 | 600 | 600 | 611 | 602 | 621 | 606 | 603 | 603
Participants
  207078_BF_Nouna: number analyzed (Participants) | 606 | 600 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207078_BF_Nouna: Male, Infected | 199 | 251 | 172 | 132 |  |  |  |  |  |
  207078_BF_Nouna: Female, Infected | 204 | 237 | 180 | 125 |  |  |  |  |  |
  207078_BF_Nouna: Male, Not infected | 103 | 49 | 120 | 188 |  |  |  |  |  |
  207078_BF_Nouna: Female, Not infected | 100 | 63 | 128 | 155 |  |  |  |  |  |
  207079_BF_Sapone: number analyzed (Participants) | 604 | 599 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207079_BF_Sapone: Male, Infected | 160 | 162 | 108 | 108 |  |  |  |  |  |
  207079_BF_Sapone: Female, Infected | 139 | 154 | 86 | 96 |  |  |  |  |  |
  207079_BF_Sapone: Male, Not infected | 149 | 154 | 204 | 200 |  |  |  |  |  |
  207079_BF_Sapone: Female, Not infected | 156 | 129 | 202 | 196 |  |  |  |  |  |
  207080_SN_Niakhar: number analyzed (Participants) | 598 | 601 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207080_SN_Niakhar: Male, Infected | 4 | 2 |  |  |  |  |  |  |  |
  207080_SN_Niakhar: Female, Infected | 5 | 1 |  |  |  |  |  |  |  |
  207080_SN_Niakhar: Male, Not infected | 285 | 319 |  |  |  |  |  |  |  |
  207080_SN_Niakhar: Female, Not infected | 304 | 279 |  |  |  |  |  |  |  |
  207081_TZ_Korogwe: number analyzed (Participants) | 601 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207081_TZ_Korogwe: Male, Infected | 32 | 9 |  |  |  |  |  |  |  |
  207081_TZ_Korogwe: Female, Infected | 31 | 9 |  |  |  |  |  |  |  |
  207081_TZ_Korogwe: Male, Not infected | 287 | 285 |  |  |  |  |  |  |  |
  207081_TZ_Korogwe: Female, Not infected | 251 | 297 |  |  |  |  |  |  |  |
  207082_KE_Kombewa: number analyzed (Participants) | 599 | 599 | 599 | 600 | 600 | 600 | 600 | 600 | 600 | 600
  207082_KE_Kombewa: Male, Infected | 106 | 95 | 111 | 105 | 101 | 89 | 68 | 67 | 80 | 54
  207082_KE_Kombewa: Female, Infected | 90 | 94 | 102 | 106 | 86 | 96 | 66 | 56 | 44 | 64
  207082_KE_Kombewa: Male, Not infected | 214 | 189 | 177 | 186 | 216 | 199 | 220 | 221 | 242 | 232
  207082_KE_Kombewa: Female, Not infected | 189 | 221 | 209 | 203 | 197 | 216 | 246 | 256 | 234 | 250
  207083_GH_Kintampo: number analyzed (Participants) | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207083_GH_Kintampo: Male, Infected | 118 | 111 |  |  |  |  |  |  |  |
  207083_GH_Kintampo: Female, Infected | 96 | 101 |  |  |  |  |  |  |  |
  207083_GH_Kintampo: Male, Not infected | 204 | 192 |  |  |  |  |  |  |  |
  207083_GH_Kintampo: Female, Not infected | 182 | 196 |  |  |  |  |  |  |  |
  207083_GH_Kintampo_EXP: number analyzed (Participants) | 0 | 0 | 600 | 600 | 600 | 600 | 600 | 600 | 600 | 600
  207083_GH_Kintampo_EXP: Male, Infected |  |  | 130 | 109 | 72 | 64 | 49 | 35 | 28 | 28
  207083_GH_Kintampo_EXP: Female, Infected |  |  | 95 | 77 | 81 | 55 | 54 | 39 | 35 | 24
  207083_GH_Kintampo_EXP: Male, Not infected |  |  | 186 | 213 | 240 | 249 | 243 | 256 | 258 | 285
  207083_GH_Kintampo_EXP: Female, Not infected |  |  | 189 | 201 | 207 | 232 | 254 | 270 | 279 | 263
  207083_GH_Kintampo_UNEXP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  207083_GH_Kintampo_UNEXP: Male, Infected |  |  |  |  |  | 86 | 63 | 47 | 48 | 37
  207083_GH_Kintampo_UNEXP: Female, Infected |  |  |  |  |  | 69 | 70 | 52 | 43 | 30
  207083_GH_Kintampo_UNEXP: Male, Not infected |  |  |  |  |  | 215 | 227 | 253 | 276 | 285
  207083_GH_Kintampo_UNEXP: Female, Not infected |  |  |  |  |  | 230 | 240 | 248 | 233 | 248
  207084_SN_Keur Soce: number analyzed (Participants) | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207084_SN_Keur Soce: Male, Infected | 1 | 5 |  |  |  |  |  |  |  |
  207084_SN_Keur Soce: Female, Infected | 2 | 1 |  |  |  |  |  |  |  |
  207084_SN_Keur Soce: Male, Not infected | 296 | 288 |  |  |  |  |  |  |  |
  207084_SN_Keur Soce: Female, Not infected | 301 | 306 |  |  |  |  |  |  |  |
  228607_GH_Navrongo_EXP: number analyzed (Participants) | 0 | 0 | 0 | 600 | 605 | 599 | 600 | 599 | 600 | 600
  228607_GH_Navrongo_EXP: Male, Infected |  |  |  | 57 | 56 | 50 | 46 | 29 | 33 | 37
  228607_GH_Navrongo_EXP: Female, Infected |  |  |  | 43 | 54 | 47 | 31 | 40 | 41 | 37
  228607_GH_Navrongo_EXP: Male, Not infected |  |  |  | 256 | 266 | 257 | 253 | 268 | 270 | 251
  228607_GH_Navrongo_EXP: Female, Not infected |  |  |  | 244 | 229 | 245 | 270 | 262 | 256 | 275
  228607_GH_Navrongo_UNEXP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  228607_GH_Navrongo_UNEXP: Male, Infected |  |  |  |  |  | 49 | 56 | 43 | 50 | 46
  228607_GH_Navrongo_UNEXP: Female, Infected |  |  |  |  |  | 57 | 39 | 32 | 39 | 49
  228607_GH_Navrongo_UNEXP: Male, Not infected |  |  |  |  |  | 270 | 260 | 265 | 279 | 259
  228607_GH_Navrongo_UNEXP: Female, Not infected |  |  |  |  |  | 224 | 245 | 260 | 232 | 246
  233149_MA_Mangochi: number analyzed (Participants) | 0 | 0 | 0 | 0 | 597 | 602 | 599 | 600 | 601 | 601
  233149_MA_Mangochi: Male, Infected |  |  |  |  | 57 | 48 | 31 | 44 | 42 | 39
  233149_MA_Mangochi: Female, Infected |  |  |  |  | 41 | 38 | 20 | 34 | 33 | 25
  233149_MA_Mangochi: Male, Not infected |  |  |  |  | 226 | 243 | 274 | 244 | 272 | 253
  233149_MA_Mangochi: Female, Not infected |  |  |  |  | 273 | 273 | 274 | 278 | 254 | 284
  233150_MA_Chikwawa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 583 | 0 | 621 | 600 | 600 | 597
  233150_MA_Chikwawa: Male, Infected |  |  |  |  | 34 |  | 51 | 18 | 12 | 18
  233150_MA_Chikwawa: Female, Infected |  |  |  |  | 35 |  | 46 | 14 | 5 | 7
  233150_MA_Chikwawa: Male, Not infected |  |  |  |  | 237 |  | 252 | 294 | 281 | 312
  233150_MA_Chikwawa: Female, Not infected |  |  |  |  | 277 |  | 272 | 274 | 302 | 260
  233149_MA_Monkey Bay: number analyzed (Participants) | 0 | 0 | 0 | 0 | 598 | 600 | 600 | 600 | 599 | 599
  233149_MA_Monkey Bay: Male, Infected |  |  |  |  | 33 | 19 | 15 | 19 | 20 | 22
  233149_MA_Monkey Bay: Female, Infected |  |  |  |  | 30 | 16 | 19 | 19 | 24 | 26
  233149_MA_Monkey Bay: Male, Not infected |  |  |  |  | 281 | 272 | 296 | 253 | 286 | 276
  233149_MA_Monkey Bay: Female, Not infected |  |  |  |  | 254 | 293 | 270 | 309 | 269 | 275
  233150_MA_St Monfort: number analyzed (Participants) | 0 | 0 | 0 | 0 | 584 | 0 | 613 | 600 | 600 | 603
  233150_MA_St Monfort: Male, Infected |  |  |  |  | 20 |  | 22 | 9 | 1 | 2
  233150_MA_St Monfort: Female, Infected |  |  |  |  | 18 |  | 31 | 5 | 1 | 2
  233150_MA_St Monfort: Male, Not infected |  |  |  |  | 277 |  | 288 | 284 | 332 | 303
  233150_MA_St Monfort: Female, Not infected |  |  |  |  | 269 |  | 272 | 302 | 266 | 296
  235578_KE_Bondo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 611 | 598 | 604 | 606 | 603 | 600
  235578_KE_Bondo: Male, Infected |  |  |  |  | 91 | 92 | 80 | 67 | 48 | 44
  235578_KE_Bondo: Female, Infected |  |  |  |  | 67 | 87 | 59 | 60 | 57 | 42
  235578_KE_Bondo: Male, Not infected |  |  |  |  | 247 | 213 | 214 | 217 | 251 | 244
  235578_KE_Bondo: Female, Not infected |  |  |  |  | 206 | 206 | 251 | 262 | 247 | 270
  235578_KE_Gem: number analyzed (Participants) | 0 | 0 | 0 | 0 | 599 | 588 | 604 | 606 | 600 | 602
  235578_KE_Gem: Male, Infected |  |  |  |  | 78 | 69 | 56 | 55 | 53 | 45
  235578_KE_Gem: Female, Infected |  |  |  |  | 68 | 62 | 59 | 51 | 57 | 43
  235578_KE_Gem: Male, Not infected |  |  |  |  | 221 | 226 | 248 | 260 | 236 | 254
  235578_KE_Gem: Female, Not infected |  |  |  |  | 232 | 231 | 241 | 240 | 254 | 260
  235579_KE_Nyando: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 606 | 600 | 600
  235579_KE_Nyando: Male, Infected |  |  |  |  |  | 88 | 51 | 42 | 57 | 44
  235579_KE_Nyando: Female, Infected |  |  |  |  |  | 65 | 56 | 32 | 37 | 45
  235579_KE_Nyando: Male, Not infected |  |  |  |  |  | 227 | 253 | 267 | 243 | 239
  235579_KE_Nyando: Female, Not infected |  |  |  |  |  | 220 | 240 | 265 | 263 | 272

3. Secondary Outcome: Number of Participants Infected With Plasmodium Species Other Than P. Falciparum
Description: The infections with other Plasmodium species were determined using a blood smear slide and microscopy. The number of participants infected with P. malaria, P. vivax and P. ovale was summarized.
Time Frame: At Day 1 (survey completion visit)
Population: The analysis was performed on the ATP Cohort which included all participants who met the eligibility criteria, adhered to the procedures defined in the protocol, had no elimination criteria during the study, had at least one laboratory result from a blood sample available and with usable data for the specified analysis at the specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group
Number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
Participants
  P. malaria | 62 | 128 | 58 | 57 | 39 | 87 | 83 | 34 | 50 | 61
  P. vivax | 0 | 1 | 8 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  P. ovale | 23 | 10 | 18 | 21 | 21 | 52 | 20 | 9 | 32 | 14

4. Secondary Outcome: Number of Participants Who Received Dose 3 of the Diphtheria, Tetanus, Pertussis/ Hepatitis B/ Haemophilus Influenzae Type b (DTP/HepB/Hib) Vaccine or Dose 1 of the Measles Vaccine
Time Frame: At Day 1 (survey completion visit)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group
Number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
Participants
  DTP/HepB/Hib [3rd dose] | 2922 | 3688 | 2029 | 2728 | 5165 | 5562 | 6745 | 6843 | 6856 | 6997
  Measles [1st dose] | 2261 | 3376 | 1897 | 2535 | 4787 | 5218 | 5435 | 6317 | 6340 | 6413

5. Secondary Outcome: Number of Participants Who Received Anti-malarial Therapy or Any Other Medication Within 14 Days Prior to the Study Visit
Description: The number of participants who received anti-malarial therapy out of those who reported malaria in the last 14 days prior to the study visit was summarized.
Time Frame: Up to 14 days prior to the study visit at Day 1
Population: The analysis was performed on the ATP Cohort which included all participants who met the eligibility criteria, adhered to the procedures defined in the protocol, had no elimination criteria during the study, had at least one laboratory result from a blood sample available and with usable data for the specified analysis for the specified time period.
Measure: Count of Participants; unit: Participants
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group
Number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 1295 | 5987 | 7241 | 7217 | 7203 | 7202
Participants | 700 | 672 | 455 | 661 | 1295 | 1041 | 783 | 769 | 1043 | 516

6. Secondary Outcome: Number of Participants With Measured Fever at the Time of Their Study Visit
Description: Fever was defined as an axillary temperature of 37.5°C or higher.
Time Frame: At Day 1 (survey completion visit)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group
Number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
Participants | 215 | 200 | 94 | 127 | 245 | 223 | 161 | 200 | 250 | 212

7. Secondary Outcome: Number of Participants With Reported Fever in the 24 Hours Prior to Their Study Visit
Description: Fever was defined as an axillary temperature of 37.5°C or higher.
Time Frame: Up to 24 hours prior to their study visit at Day 1
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group
Number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
Participants | 1060 | 1082 | 624 | 822 | 1307 | 1162 | 1133 | 1072 | 1235 | 1099

8. Secondary Outcome: Number of Participants Demonstrating Care-seeking Behavior Following Reported Fever or Malaria up to 14 Days Prior to Their Study Visit
Description: The number of participants demonstrating care-seeking behavior following reported fever or malaria was summarized by where the participant was taken for treatment (home, drug seller, pharmacy, private clinic, health center, hospital, other, not applicable [no treatment received]), by when the participant was taken for treatment (at onset, when the participant did not improve, when the participant got worse, other, not applicable [no treatment received], missing [participant was taken for treatment but did not answer the question regarding when]) and by what time the participant was taken for treatment (the same day, the next day, 2 days later, more than 2 days later, not applicable [no treatment received], missing [participant was taken for treatment but did not answer the question regarding the time]).
Time Frame: Up to 14 days prior to their study visit at Day 1
Population: The analysis was performed on the ATP Cohort which included all participants who met the eligibility criteria, adhered to the procedures defined in the protocol, had no elimination criteria during the study, had at least one laboratory result from a blood sample available and with usable data for the specified analysis for the specified time period. Here, 'number analyzed' = participants with available data for each specified row.
Measure: Count of Participants; unit: Participants
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group
Number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
Participants
  Where the participant was taken for treatment - Home | 117 | 102 | 42 | 88 | 209 | 194 | 130 | 94 | 208 | 110
  Where the participant was taken for treatment - Drug seller | 94 | 163 | 152 | 109 | 149 | 172 | 158 | 111 | 153 | 77
  Where the participant was taken for treatment - Pharmacy | 97 | 45 | 11 | 48 | 135 | 124 | 101 | 106 | 111 | 73
  Where the participant was taken for treatment - Private clinic | 26 | 24 | 20 | 10 | 68 | 44 | 23 | 47 | 25 | 26
  Where the participant was taken for treatment - Health center | 196 | 146 | 105 | 255 | 392 | 299 | 238 | 237 | 302 | 156
  Where the participant was taken for treatment - Hospital | 40 | 40 | 31 | 46 | 77 | 67 | 53 | 66 | 50 | 26
  Where the participant was taken for treatment - Other | 86 | 17 | 1 | 10 | 77 | 108 | 20 | 47 | 48 | 34
  Where the participant was taken for treatment - Not Applicable | 3546 | 3662 | 2037 | 2429 | 4267 | 4977 | 6516 | 6509 | 6306 | 6700
  Where the participant was taken for treatment - Missing: number analyzed (Participants) | 4208 | 0 | 0 | 3000 | 5377 | 5987 | 7241 | 0 | 0 | 0
  Where the participant was taken for treatment - Missing | 6 |  |  | 5 | 3 | 2 | 2 |  |  |
  When the participant was taken for treatment - At onset | 358 | 355 | 323 | 477 | 707 | 651 | 520 | 525 | 686 | 356
  When the participant was taken for treatment - When participant did not improve | 33 | 23 | 29 | 86 | 346 | 263 | 178 | 145 | 159 | 118
  When the participant was taken for treatment - When participant got worse | 11 | 5 | 7 | 7 | 43 | 92 | 26 | 35 | 52 | 28
  When the participant was taken for treatment - Other | 49 | 1 | 0 | 0 | 5 | 1 | 0 | 1 | 0 | 0
  When the participant was taken for treatment - Not Applicable | 3546 | 3662 | 2037 | 2429 | 4267 | 4977 | 6516 | 6509 | 6306 | 6700
  When the participant was taken for treatment - Missing: number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 0 | 0
  When the participant was taken for treatment - Missing | 211 | 153 | 3 | 1 | 3 | 3 | 1 | 2 |  |
  What time the participant was taken for treatment - Same day | 300 | 278 | 213 | 416 | 707 | 610 | 473 | 464 | 596 | 310
  What time the participant was taken for treatment - Next day | 59 | 83 | 121 | 127 | 346 | 258 | 177 | 172 | 239 | 151
  What time the participant was taken for treatment - Two days later | 28 | 11 | 17 | 17 | 43 | 71 | 53 | 43 | 38 | 29
  What time the participant was taken for treatment - More than 2 days later | 29 | 11 | 9 | 6 | 5 | 65 | 20 | 26 | 23 | 12
  What time the participant was taken for treatment - Not Applicable | 3546 | 3662 | 2037 | 2429 | 4267 | 4977 | 6516 | 6509 | 6306 | 6700
  What time the participant was taken for treatment - Missing: number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 0
  What time the participant was taken for treatment - Missing | 246 | 154 | 2 | 5 | 17 | 6 | 2 | 3 | 1 |

9. Secondary Outcome: Number of Participants in Each Geo-referenced Segment
Description: The number of participants was summarized by: center number/ country [BF, SN, TZ, KE, GH, MA]/ city followed by the segment ID. Positioning of the participant's residence was attributed to a segment with a unique ID from the grid referencing study area map in which the participant resided; where necessary, grouping small geographically proximate villages so that each segment had at least 10 study participants to avoid personally identifiable information (PII), and proceeding as far as geographically appropriate.
Time Frame: At Day 1 (survey completion visit)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group
Number analyzed (Participants) | 606 | 601 | 600 | 600 | 611 | 602 | 621 | 606 | 603 | 603
Participants
  207078_BF_Nouna, ID-20707860: number analyzed (Participants) | 606 | 600 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207078_BF_Nouna, ID-20707860 | 21 | 58 | 11 | 30 |  |  |  |  |  |
  207078_BF_Nouna, ID-20707861: number analyzed (Participants) | 606 | 600 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207078_BF_Nouna, ID-20707861 | 50 | 66 | 55 | 38 |  |  |  |  |  |
  207078_BF_Nouna, ID-20707862: number analyzed (Participants) | 606 | 600 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207078_BF_Nouna, ID-20707862 | 21 | 26 | 20 | 31 |  |  |  |  |  |
  207078_BF_Nouna, ID-20707863: number analyzed (Participants) | 606 | 600 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207078_BF_Nouna, ID-20707863 | 38 | 26 | 37 | 27 |  |  |  |  |  |
  207078_BF_Nouna, ID-20707864: number analyzed (Participants) | 606 | 600 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207078_BF_Nouna, ID-20707864 | 27 | 77 | 39 | 33 |  |  |  |  |  |
  207078_BF_Nouna, ID-20707865: number analyzed (Participants) | 606 | 600 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207078_BF_Nouna, ID-20707865 | 39 | 45 | 48 | 53 |  |  |  |  |  |
  207078_BF_Nouna, ID-20707866: number analyzed (Participants) | 606 | 600 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207078_BF_Nouna, ID-20707866 | 38 | 233 | 51 | 27 |  |  |  |  |  |
  207078_BF_Nouna, ID-20707867: number analyzed (Participants) | 606 | 600 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207078_BF_Nouna, ID-20707867 | 23 | 27 | 22 | 34 |  |  |  |  |  |
  207078_BF_Nouna, ID-20707868: number analyzed (Participants) | 606 | 600 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207078_BF_Nouna, ID-20707868 | 218 | 42 | 178 | 172 |  |  |  |  |  |
  207078_BF_Nouna, ID-20707869: number analyzed (Participants) | 606 | 0 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207078_BF_Nouna, ID-20707869 | 18 |  | 16 | 24 |  |  |  |  |  |
  207078_BF_Nouna, ID-20707870: number analyzed (Participants) | 606 | 0 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207078_BF_Nouna, ID-20707870 | 23 |  | 40 | 22 |  |  |  |  |  |
  207078_BF_Nouna, ID-20707871: number analyzed (Participants) | 606 | 0 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207078_BF_Nouna, ID-20707871 | 30 |  | 25 | 39 |  |  |  |  |  |
  207078_BF_Nouna, ID-20707872: number analyzed (Participants) | 606 | 0 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207078_BF_Nouna, ID-20707872 | 28 |  | 40 | 44 |  |  |  |  |  |
  207078_BF_Nouna, ID-20707873: number analyzed (Participants) | 606 | 0 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207078_BF_Nouna, ID-20707873 | 32 |  | 18 | 26 |  |  |  |  |  |
  207079_BF_Sapone, ID-1: number analyzed (Participants) | 604 | 599 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207079_BF_Sapone, ID-1 | 57 | 51 | 69 | 70 |  |  |  |  |  |
  207079_BF_Sapone, ID-10: number analyzed (Participants) | 604 | 599 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207079_BF_Sapone, ID-10 | 65 | 69 | 64 | 52 |  |  |  |  |  |
  207079_BF_Sapone, ID-11: number analyzed (Participants) | 604 | 599 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207079_BF_Sapone, ID-11 | 34 | 25 | 25 | 19 |  |  |  |  |  |
  207079_BF_Sapone, ID-12: number analyzed (Participants) | 604 | 599 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207079_BF_Sapone, ID-12 | 13 | 34 | 28 | 40 |  |  |  |  |  |
  207079_BF_Sapone, ID-13: number analyzed (Participants) | 604 | 599 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207079_BF_Sapone, ID-13 | 29 | 48 | 46 | 43 |  |  |  |  |  |
  207079_BF_Sapone, ID-14: number analyzed (Participants) | 604 | 599 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207079_BF_Sapone, ID-14 | 15 | 26 | 32 | 33 |  |  |  |  |  |
  207079_BF_Sapone, ID-2: number analyzed (Participants) | 604 | 599 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207079_BF_Sapone, ID-2 | 45 | 41 | 41 | 37 |  |  |  |  |  |
  207079_BF_Sapone, ID-3: number analyzed (Participants) | 604 | 599 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207079_BF_Sapone, ID-3 | 42 | 39 | 53 | 58 |  |  |  |  |  |
  207079_BF_Sapone, ID-4: number analyzed (Participants) | 604 | 599 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207079_BF_Sapone, ID-4 | 59 | 48 | 57 | 67 |  |  |  |  |  |
  207079_BF_Sapone, ID-5: number analyzed (Participants) | 604 | 599 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207079_BF_Sapone, ID-5 | 47 | 45 | 38 | 45 |  |  |  |  |  |
  207079_BF_Sapone, ID-6: number analyzed (Participants) | 604 | 599 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207079_BF_Sapone, ID-6 | 40 | 49 | 41 | 34 |  |  |  |  |  |
  207079_BF_Sapone, ID-7: number analyzed (Participants) | 604 | 599 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207079_BF_Sapone, ID-7 | 45 | 36 | 34 | 28 |  |  |  |  |  |
  207079_BF_Sapone, ID-8: number analyzed (Participants) | 604 | 599 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207079_BF_Sapone, ID-8 | 78 | 51 | 44 | 53 |  |  |  |  |  |
  207079_BF_Sapone, ID-9: number analyzed (Participants) | 604 | 599 | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0
  207079_BF_Sapone, ID-9 | 35 | 37 | 28 | 21 |  |  |  |  |  |
  207080_SN_Niakhar, ID-1: number analyzed (Participants) | 598 | 601 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207080_SN_Niakhar, ID-1 | 32 | 51 |  |  |  |  |  |  |  |
  207080_SN_Niakhar, ID-2: number analyzed (Participants) | 598 | 601 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207080_SN_Niakhar, ID-2 | 69 | 106 |  |  |  |  |  |  |  |
  207080_SN_Niakhar, ID-3: number analyzed (Participants) | 598 | 601 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207080_SN_Niakhar, ID-3 | 50 | 54 |  |  |  |  |  |  |  |
  207080_SN_Niakhar, ID-4: number analyzed (Participants) | 598 | 601 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207080_SN_Niakhar, ID-4 | 49 | 33 |  |  |  |  |  |  |  |
  207080_SN_Niakhar, ID-5: number analyzed (Participants) | 598 | 601 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207080_SN_Niakhar, ID-5 | 89 | 93 |  |  |  |  |  |  |  |
  207080_SN_Niakhar, ID-6: number analyzed (Participants) | 598 | 601 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207080_SN_Niakhar, ID-6 | 19 | 19 |  |  |  |  |  |  |  |
  207080_SN_Niakhar, ID-7: number analyzed (Participants) | 598 | 601 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207080_SN_Niakhar, ID-7 | 104 | 75 |  |  |  |  |  |  |  |
  207080_SN_Niakhar, ID-8: number analyzed (Participants) | 598 | 601 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207080_SN_Niakhar, ID-8 | 94 | 87 |  |  |  |  |  |  |  |
  207080_SN_Niakhar, ID-9: number analyzed (Participants) | 598 | 601 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207080_SN_Niakhar, ID-9 | 92 | 83 |  |  |  |  |  |  |  |
  207081_TZ_Korogwe, ID-1: number analyzed (Participants) | 601 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207081_TZ_Korogwe, ID-1 | 17 | 27 |  |  |  |  |  |  |  |
  207081_TZ_Korogwe, ID-2: number analyzed (Participants) | 601 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207081_TZ_Korogwe, ID-2 | 135 | 130 |  |  |  |  |  |  |  |
  207081_TZ_Korogwe, ID-3: number analyzed (Participants) | 601 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207081_TZ_Korogwe, ID-3 | 83 | 108 |  |  |  |  |  |  |  |
  207081_TZ_Korogwe, ID-4: number analyzed (Participants) | 601 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207081_TZ_Korogwe, ID-4 | 132 | 138 |  |  |  |  |  |  |  |
  207081_TZ_Korogwe, ID-5: number analyzed (Participants) | 601 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207081_TZ_Korogwe, ID-5 | 42 | 42 |  |  |  |  |  |  |  |
  207081_TZ_Korogwe, ID-6: number analyzed (Participants) | 601 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207081_TZ_Korogwe, ID-6 | 77 | 61 |  |  |  |  |  |  |  |
  207081_TZ_Korogwe, ID-7: number analyzed (Participants) | 601 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207081_TZ_Korogwe, ID-7 | 115 | 94 |  |  |  |  |  |  |  |
  207082_KE_Kombewa, ID-11: number analyzed (Participants) | 599 | 599 | 599 | 600 | 600 | 600 | 600 | 600 | 600 | 600
  207082_KE_Kombewa, ID-11 | 140 | 75 | 133 | 129 | 133 | 120 | 118 | 112 | 79 | 146
  207082_KE_Kombewa, ID-12: number analyzed (Participants) | 599 | 599 | 599 | 600 | 600 | 600 | 600 | 600 | 600 | 600
  207082_KE_Kombewa, ID-12 | 31 | 52 | 48 | 47 | 42 | 66 | 51 | 66 | 89 | 54
  207082_KE_Kombewa, ID-13: number analyzed (Participants) | 599 | 599 | 599 | 600 | 600 | 600 | 600 | 600 | 600 | 600
  207082_KE_Kombewa, ID-13 | 82 | 68 | 58 | 69 | 82 | 57 | 63 | 59 | 148 | 85
  207082_KE_Kombewa, ID-14: number analyzed (Participants) | 599 | 599 | 599 | 600 | 600 | 600 | 600 | 600 | 600 | 600
  207082_KE_Kombewa, ID-14 | 54 | 29 | 44 | 57 | 45 | 39 | 67 | 30 | 61 | 49
  207082_KE_Kombewa, ID-21: number analyzed (Participants) | 599 | 599 | 599 | 600 | 600 | 600 | 600 | 600 | 600 | 600
  207082_KE_Kombewa, ID-21 | 58 | 75 | 65 | 100 | 68 | 68 | 90 | 79 | 57 | 71
  207082_KE_Kombewa, ID-22: number analyzed (Participants) | 599 | 599 | 599 | 600 | 600 | 600 | 600 | 600 | 600 | 600
  207082_KE_Kombewa, ID-22 | 91 | 124 | 109 | 68 | 83 | 79 | 34 | 51 | 8 | 77
  207082_KE_Kombewa, ID-23: number analyzed (Participants) | 599 | 599 | 599 | 600 | 600 | 600 | 600 | 600 | 600 | 600
  207082_KE_Kombewa, ID-23 | 54 | 104 | 74 | 54 | 65 | 70 | 65 | 126 | 72 | 59
  207082_KE_Kombewa, ID-24: number analyzed (Participants) | 599 | 599 | 599 | 600 | 600 | 600 | 600 | 600 | 600 | 600
  207082_KE_Kombewa, ID-24 | 89 | 72 | 68 | 76 | 82 | 101 | 112 | 77 | 86 | 59
  207083_GH_Kintampo, ID-1: number analyzed (Participants) | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207083_GH_Kintampo, ID-1 | 163 | 158 |  |  |  |  |  |  |  |
  207083_GH_Kintampo, ID-2: number analyzed (Participants) | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207083_GH_Kintampo, ID-2 | 257 | 168 |  |  |  |  |  |  |  |
  207083_GH_Kintampo, ID-3: number analyzed (Participants) | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207083_GH_Kintampo, ID-3 | 180 | 274 |  |  |  |  |  |  |  |
  207084_SN_Keur Soce, ID-1: number analyzed (Participants) | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207084_SN_Keur Soce, ID-1 | 148 | 139 |  |  |  |  |  |  |  |
  207084_SN_Keur Soce, ID-2: number analyzed (Participants) | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207084_SN_Keur Soce, ID-2 | 243 | 269 |  |  |  |  |  |  |  |
  207084_SN_Keur Soce, ID-3: number analyzed (Participants) | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207084_SN_Keur Soce, ID-3 | 142 | 136 |  |  |  |  |  |  |  |
  207084_SN_Keur Soce, ID-4: number analyzed (Participants) | 600 | 600 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  207084_SN_Keur Soce, ID-4 | 67 | 56 |  |  |  |  |  |  |  |
  207083_GH_Kintampo_EXP, ID-1: number analyzed (Participants) | 0 | 0 | 600 | 600 | 600 | 600 | 600 | 600 | 600 | 600
  207083_GH_Kintampo_EXP, ID-1 |  |  | 188 | 250 | 248 | 359 | 276 | 266 | 335 | 299
  207083_GH_Kintampo_EXP, ID-2: number analyzed (Participants) | 0 | 0 | 600 | 600 | 600 | 600 | 600 | 600 | 600 | 600
  207083_GH_Kintampo_EXP, ID-2 |  |  | 242 | 207 | 213 | 160 | 214 | 246 | 180 | 167
  207083_GH_Kintampo_EXP, ID-3: number analyzed (Participants) | 0 | 0 | 600 | 600 | 600 | 600 | 600 | 600 | 600 | 600
  207083_GH_Kintampo_EXP, ID-3 |  |  | 170 | 143 | 139 | 81 | 110 | 88 | 85 | 134
  207083_GH_Kintampo_UNEXP, ID-2070831: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  207083_GH_Kintampo_UNEXP, ID-2070831 |  |  |  |  |  | 130 | 130 | 151 | 164 | 179
  207083_GH_Kintampo_UNEXP, ID-2070832: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  207083_GH_Kintampo_UNEXP, ID-2070832 |  |  |  |  |  | 296 | 287 | 268 | 269 | 229
  207083_GH_Kintampo_UNEXP, ID-2070833: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  207083_GH_Kintampo_UNEXP, ID-2070833 |  |  |  |  |  | 174 | 183 | 181 | 167 | 192
  228607_GH_Navrongo_EXP, ID-2286071: number analyzed (Participants) | 0 | 0 | 0 | 600 | 605 | 599 | 600 | 599 | 600 | 600
  228607_GH_Navrongo_EXP, ID-2286071 |  |  |  | 41 | 56 | 78 | 94 | 55 | 39 | 124
  228607_GH_Navrongo_EXP, ID-2286072: number analyzed (Participants) | 0 | 0 | 0 | 600 | 605 | 599 | 600 | 599 | 600 | 600
  228607_GH_Navrongo_EXP, ID-2286072 |  |  |  | 110 | 133 | 124 | 88 | 103 | 120 | 136
  228607_GH_Navrongo_EXP, ID-2286073: number analyzed (Participants) | 0 | 0 | 0 | 600 | 605 | 599 | 600 | 599 | 600 | 600
  228607_GH_Navrongo_EXP, ID-2286073 |  |  |  | 127 | 108 | 125 | 118 | 162 | 124 | 162
  228607_GH_Navrongo_EXP, ID-2286074: number analyzed (Participants) | 0 | 0 | 0 | 600 | 605 | 599 | 600 | 599 | 600 | 600
  228607_GH_Navrongo_EXP, ID-2286074 |  |  |  | 188 | 190 | 168 | 191 | 172 | 224 | 83
  228607_GH_Navrongo_EXP, ID-2286075: number analyzed (Participants) | 0 | 0 | 0 | 600 | 605 | 599 | 600 | 599 | 600 | 600
  228607_GH_Navrongo_EXP, ID-2286075 |  |  |  | 134 | 118 | 93 | 109 | 107 | 93 | 95
  228607_GH_Navrongo_EXP, ID-22860705: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 599 | 0 | 0 | 0 | 0
  228607_GH_Navrongo_EXP, ID-22860705 |  |  |  |  |  | 10 |  |  |  |
  228607_GH_Navrongo_EXP, ID-22860712: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 599 | 0 | 0 | 0 | 0
  228607_GH_Navrongo_EXP, ID-22860712 |  |  |  |  |  | 124 |  |  |  |
  228607_GH_Navrongo_UNEXP, ID-22860709: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 0 | 0 | 0 | 0
  228607_GH_Navrongo_UNEXP, ID-22860709 |  |  |  |  |  | 8 |  |  |  |
  228607_GH_Navrongo_UNEXP, ID-2286071: number analyzed (Participants) | 0 | 00 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  228607_GH_Navrongo_UNEXP, ID-2286071 |  |  |  |  |  | 10 | 9 | 11 | 9 | 13
  228607_GH_Navrongo_UNEXP, ID-22860710: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  228607_GH_Navrongo_UNEXP, ID-22860710 |  |  |  |  |  | 52 | 29 | 18 | 38 | 43
  228607_GH_Navrongo_UNEXP, ID-22860711: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  228607_GH_Navrongo_UNEXP, ID-22860711 |  |  |  |  |  | 32 | 33 | 22 | 41 | 36
  228607_GH_Navrongo_UNEXP, ID-22860712: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  228607_GH_Navrongo_UNEXP, ID-22860712 |  |  |  |  |  | 89 | 90 | 80 | 75 | 75
  228607_GH_Navrongo_UNEXP, ID-22860713: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  228607_GH_Navrongo_UNEXP, ID-22860713 |  |  |  |  |  | 15 | 12 | 2 | 12 | 7
  228607_GH_Navrongo_UNEXP, ID-22860714: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  228607_GH_Navrongo_UNEXP, ID-22860714 |  |  |  |  |  | 3 | 3 | 2 | 20 | 7
  228607_GH_Navrongo_UNEXP, ID-2286072: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  228607_GH_Navrongo_UNEXP, ID-2286072 |  |  |  |  |  | 66 | 70 | 67 | 70 | 63
  228607_GH_Navrongo_UNEXP, ID-2286073: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  228607_GH_Navrongo_UNEXP, ID-2286073 |  |  |  |  |  | 18 | 18 | 14 | 11 | 18
  228607_GH_Navrongo_UNEXP, ID-2286074: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  228607_GH_Navrongo_UNEXP, ID-2286074 |  |  |  |  |  | 80 | 91 | 82 | 104 | 84
  228607_GH_Navrongo_UNEXP, ID-2286075: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  228607_GH_Navrongo_UNEXP, ID-2286075 |  |  |  |  |  | 12 | 9 | 9 | 6 | 9
  228607_GH_Navrongo_UNEXP, ID-2286076: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  228607_GH_Navrongo_UNEXP, ID-2286076 |  |  |  |  |  | 12 | 38 | 46 | 37 | 25
  228607_GH_Navrongo_UNEXP, ID-2286077: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  228607_GH_Navrongo_UNEXP, ID-2286077 |  |  |  |  |  | 46 | 43 | 39 | 48 | 39
  228607_GH_Navrongo_UNEXP, ID-2286078: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  228607_GH_Navrongo_UNEXP, ID-2286078 |  |  |  |  |  | 60 | 53 | 77 | 26 | 50
  228607_GH_Navrongo_UNEXP, ID-2286079: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 600 | 600 | 600
  228607_GH_Navrongo_UNEXP, ID-2286079 |  |  |  |  |  | 97 | 102 | 131 | 103 | 131
  233149_MA_Mangochi, ID-23314902: number analyzed (Participants) | 0 | 0 | 0 | 0 | 597 | 0 | 0 | 0 | 0 | 0
  233149_MA_Mangochi, ID-23314902 |  |  |  |  | 1 |  |  |  |  |
  233149_MA_Mangochi, ID-23314911: number analyzed (Participants) | 0 | 0 | 0 | 0 | 597 | 602 | 599 | 600 | 601 | 601
  233149_MA_Mangochi, ID-23314911 |  |  |  |  | 143 | 239 | 240 | 279 | 254 | 187
  233149_MA_Mangochi, ID-23314912: number analyzed (Participants) | 0 | 0 | 0 | 0 | 597 | 602 | 599 | 600 | 601 | 601
  233149_MA_Mangochi, ID-23314912 |  |  |  |  | 223 | 261 | 246 | 196 | 169 | 319
  233149_MA_Mangochi, ID-23314913: number analyzed (Participants) | 0 | 0 | 0 | 0 | 597 | 602 | 599 | 600 | 601 | 601
  233149_MA_Mangochi, ID-23314913 |  |  |  |  | 214 | 102 | 113 | 125 | 177 | 92
  233149_MA_Mangochi, ID-23314921: number analyzed (Participants) | 0 | 0 | 0 | 0 | 597 | 0 | 0 | 0 | 0 | 601
  233149_MA_Mangochi, ID-23314921 |  |  |  |  | 16 |  |  |  |  | 2
  233149_MA_Mangochi, ID-23314922: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 601
  233149_MA_Mangochi, ID-23314922 |  |  |  |  |  |  |  |  |  | 1
  233149_MA_Monkey Bay, ID-23314911: number analyzed (Participants) | 0 | 0 | 0 | 0 | 598 | 600 | 0 | 0 | 0 | 0
  233149_MA_Monkey Bay, ID-23314911 |  |  |  |  | 2 | 18 |  |  |  |
  233149_MA_Monkey Bay, ID-23314912: number analyzed (Participants) | 0 | 0 | 0 | 0 | 598 | 0 | 0 | 0 | 0 | 599
  233149_MA_Monkey Bay, ID-23314912 |  |  |  |  | 1 |  |  |  |  | 3
  233149_MA_Monkey Bay, ID-23314921: number analyzed (Participants) | 0 | 0 | 0 | 0 | 598 | 600 | 600 | 600 | 599 | 599
  233149_MA_Monkey Bay, ID-23314921 |  |  |  |  | 149 | 167 | 157 | 179 | 239 | 241
  233149_MA_Monkey Bay, ID-23314922: number analyzed (Participants) | 0 | 0 | 0 | 0 | 598 | 600 | 600 | 600 | 599 | 599
  233149_MA_Monkey Bay, ID-23314922 |  |  |  |  | 446 | 410 | 443 | 421 | 360 | 355
  233149_MA_Monkey Bay, ID-23314913: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 0 | 0 | 0 | 0
  233149_MA_Monkey Bay, ID-23314913 |  |  |  |  |  | 5 |  |  |  |
  233150_MA_Chikwawa, ID-23315006: number analyzed (Participants) | 0 | 0 | 0 | 0 | 598 | 0 | 0 | 0 | 0 | 0
  233150_MA_Chikwawa, ID-23315006 |  |  |  |  | 39 |  |  |  |  |
  233150_MA_Chikwawa, ID-23315007: number analyzed (Participants) | 0 | 0 | 0 | 0 | 598 | 0 | 621 | 600 | 600 | 597
  233150_MA_Chikwawa, ID-23315007 |  |  |  |  | 53 |  | 92 | 112 | 57 | 52
  233150_MA_Chikwawa, ID-23315008: number analyzed (Participants) | 0 | 0 | 0 | 0 | 598 | 0 | 621 | 600 | 600 | 597
  233150_MA_Chikwawa, ID-23315008 |  |  |  |  | 117 |  | 55 | 225 | 228 | 228
  233150_MA_Chikwawa, ID-23315010: number analyzed (Participants) | 0 | 0 | 0 | 0 | 598 | 0 | 621 | 600 | 600 | 597
  233150_MA_Chikwawa, ID-23315010 |  |  |  |  | 292 |  | 346 | 156 | 289 | 246
  233150_MA_Chikwawa, ID-23315011: number analyzed (Participants) | 0 | 0 | 0 | 0 | 598 | 0 | 621 | 600 | 600 | 597
  233150_MA_Chikwawa, ID-23315011 |  |  |  |  | 42 |  | 42 | 88 | 21 | 69
  233150_MA_Chikwawa, ID-23315012: number analyzed (Participants) | 0 | 0 | 0 | 0 | 598 | 0 | 621 | 600 | 0 | 0
  233150_MA_Chikwawa, ID-23315012 |  |  |  |  | 40 |  | 86 | 17 |  |
  233150_MA_Chikwawa, ID-23315001: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 600 | 0 | 597
  233150_MA_Chikwawa, ID-23315001 |  |  |  |  |  |  |  | 1 |  | 2
  233150_MA_Chikwawa, ID-23315005: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 600 | 0 | 0
  233150_MA_Chikwawa, ID-23315005 |  |  |  |  |  |  |  | 1 |  |
  233150_MA_Chikwawa, ID-23315003: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 600 | 0
  233150_MA_Chikwawa, ID-23315003 |  |  |  |  |  |  |  |  | 5 |
  233150_MA_St Monfort, ID-23315001: number analyzed (Participants) | 0 | 0 | 0 | 0 | 584 | 0 | 0 | 0 | 0 | 603
  233150_MA_St Monfort, ID-23315001 |  |  |  |  | 1 |  |  |  |  | 1
  233150_MA_St Monfort, ID-23315002: number analyzed (Participants) | 0 | 0 | 0 | 0 | 584 | 0 | 613 | 600 | 600 | 603
  233150_MA_St Monfort, ID-23315002 |  |  |  |  | 13 |  | 231 | 186 | 89 | 81
  233150_MA_St Monfort, ID-23315003: number analyzed (Participants) | 0 | 0 | 0 | 0 | 584 | 0 | 613 | 600 | 600 | 603
  233150_MA_St Monfort, ID-23315003 |  |  |  |  | 14 |  | 174 | 264 | 233 | 251
  233150_MA_St Monfort, ID-23315005: number analyzed (Participants) | 0 | 0 | 0 | 0 | 584 | 0 | 613 | 600 | 600 | 603
  233150_MA_St Monfort, ID-23315005 |  |  |  |  | 10 |  | 207 | 150 | 278 | 267
  233150_MA_St Monfort, ID-23315010: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 613 | 0 | 0 | 603
  233150_MA_St Monfort, ID-23315010 |  |  |  |  |  |  | 1 |  |  | 2
  233150_MA_St Monfort, ID-23315011: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 603
  233150_MA_St Monfort, ID-23315011 |  |  |  |  |  |  |  |  |  | 1
  235578_KE_Bondo, ID-23557801: number analyzed (Participants) | 0 | 0 | 0 | 0 | 611 | 598 | 604 | 606 | 603 | 600
  235578_KE_Bondo, ID-23557801 |  |  |  |  | 108 | 80 | 49 | 64 | 69 | 67
  235578_KE_Bondo, ID-23557802: number analyzed (Participants) | 0 | 0 | 0 | 0 | 611 | 598 | 604 | 606 | 603 | 600
  235578_KE_Bondo, ID-23557802 |  |  |  |  | 85 | 131 | 128 | 145 | 123 | 137
  235578_KE_Bondo, ID-23557803: number analyzed (Participants) | 0 | 0 | 0 | 0 | 611 | 598 | 604 | 606 | 603 | 600
  235578_KE_Bondo, ID-23557803 |  |  |  |  | 147 | 99 | 113 | 110 | 105 | 106
  235578_KE_Bondo, ID-23557804: number analyzed (Participants) | 0 | 0 | 0 | 0 | 611 | 598 | 604 | 606 | 603 | 600
  235578_KE_Bondo, ID-23557804 |  |  |  |  | 115 | 63 | 119 | 122 | 119 | 114
  235578_KE_Bondo, ID-23557805: number analyzed (Participants) | 0 | 0 | 0 | 0 | 611 | 598 | 604 | 606 | 603 | 600
  235578_KE_Bondo, ID-23557805 |  |  |  |  | 101 | 79 | 96 | 79 | 88 | 92
  235578_KE_Bondo, ID-23557806: number analyzed (Participants) | 0 | 0 | 0 | 0 | 611 | 598 | 604 | 606 | 603 | 600
  235578_KE_Bondo, ID-23557806 |  |  |  |  | 55 | 146 | 99 | 86 | 99 | 84
  235578_KE_Gem, ID-23557801: number analyzed (Participants) | 0 | 0 | 0 | 0 | 599 | 588 | 604 | 606 | 600 | 602
  235578_KE_Gem, ID-23557801 |  |  |  |  | 86 | 135 | 108 | 88 | 92 | 116
  235578_KE_Gem, ID-23557802: number analyzed (Participants) | 0 | 0 | 0 | 0 | 599 | 588 | 604 | 606 | 600 | 602
  235578_KE_Gem, ID-23557802 |  |  |  |  | 83 | 52 | 90 | 112 | 112 | 100
  235578_KE_Gem, ID-23557803: number analyzed (Participants) | 0 | 0 | 0 | 0 | 599 | 588 | 604 | 606 | 600 | 602
  235578_KE_Gem, ID-23557803 |  |  |  |  | 141 | 73 | 106 | 114 | 104 | 122
  235578_KE_Gem, ID-23557804: number analyzed (Participants) | 0 | 0 | 0 | 0 | 599 | 588 | 604 | 606 | 600 | 602
  235578_KE_Gem, ID-23557804 |  |  |  |  | 124 | 93 | 99 | 114 | 129 | 123
  235578_KE_Gem, ID-23557805: number analyzed (Participants) | 0 | 0 | 0 | 0 | 599 | 588 | 604 | 606 | 600 | 602
  235578_KE_Gem, ID-23557805 |  |  |  |  | 88 | 197 | 135 | 107 | 86 | 79
  235578_KE_Gem, ID-23557806: number analyzed (Participants) | 0 | 0 | 0 | 0 | 599 | 588 | 604 | 606 | 600 | 602
  235578_KE_Gem, ID-23557806 |  |  |  |  | 77 | 38 | 66 | 71 | 77 | 62
  235579_KE_Nyando, ID-23557911: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 606 | 600 | 600
  235579_KE_Nyando, ID-23557911 |  |  |  |  |  | 60 | 55 | 59 | 80 | 146
  235579_KE_Nyando, ID-23557912: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 606 | 600 | 600
  235579_KE_Nyando, ID-23557912 |  |  |  |  |  | 48 | 69 | 54 | 48 | 104
  235579_KE_Nyando, ID-23557913: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 606 | 600 | 600
  235579_KE_Nyando, ID-23557913 |  |  |  |  |  | 42 | 55 | 54 | 46 | 81
  235579_KE_Nyando, ID-23557914: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 606 | 600 | 600
  235579_KE_Nyando, ID-23557914 |  |  |  |  |  | 23 | 19 | 34 | 39 | 75
  235579_KE_Nyando, ID-23557915: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 606 | 600 | 600
  235579_KE_Nyando, ID-23557915 |  |  |  |  |  | 28 | 37 | 31 | 42 | 75
  235579_KE_Nyando, ID-23557916: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 606 | 600 | 600
  235579_KE_Nyando, ID-23557916 |  |  |  |  |  | 86 | 61 | 62 | 74 | 55
  235579_KE_Nyando, ID-23557921: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 606 | 600 | 600
  235579_KE_Nyando, ID-23557921 |  |  |  |  |  | 7 | 16 | 23 | 9 | 10
  235579_KE_Nyando, ID-23557922: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 606 | 600 | 600
  235579_KE_Nyando, ID-23557922 |  |  |  |  |  | 64 | 53 | 27 | 33 | 10
  235579_KE_Nyando, ID-23557923: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 606 | 600 | 600
  235579_KE_Nyando, ID-23557923 |  |  |  |  |  | 54 | 39 | 47 | 37 | 6
  235579_KE_Nyando, ID-23557924: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 606 | 600 | 600
  235579_KE_Nyando, ID-23557924 |  |  |  |  |  | 17 | 11 | 19 | 37 | 19
  235579_KE_Nyando, ID-23557925: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 606 | 600 | 600
  235579_KE_Nyando, ID-23557925 |  |  |  |  |  | 20 | 26 | 35 | 28 | 2
  235579_KE_Nyando, ID-23557926: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 606 | 600 | 600
  235579_KE_Nyando, ID-23557926 |  |  |  |  |  | 46 | 46 | 32 | 41 | 4
  235579_KE_Nyando, ID-23557927: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 606 | 600 | 600
  235579_KE_Nyando, ID-23557927 |  |  |  |  |  | 46 | 85 | 68 | 51 | 13
  235579_KE_Nyando, ID-23557928: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 600 | 600 | 606 | 600 | 0
  235579_KE_Nyando, ID-23557928 |  |  |  |  |  | 59 | 28 | 61 | 35 |

10. Secondary Outcome: Number of Participants Experiencing Malaria Risk Factors Categorized by the Number of Participants Living in the Same House (by Parasite Density)
Description: Participants were categorized by the number of people living in the same house relative to enrolled participants as follows: less than of equal to (<=) 3 per 1 enrolled (LE 3/1), 4-5 per 1 (4-5/1), more than (>) 5 per 1 (GT 5/1); <=3 per 2 enrolled (LE 3/2), 4-5 per 2 (4-5/2), >5 per 2 (GT 5/2); <=3 per 3 enrolled (LE 3/3), 4-5 per 3 (4-5/3), >5 per 3 (GT 5/3); 4-5 per more than 3 enrolled (4-5/GT 3), >5 per more than 3 enrolled (GT 5/GT 3). Participants were also categorized by parasite density: low (<2500 parasites/μL), medium (2500-9999/μL), high (10000-19999/μL), very high (>=20000/μL), negative, and missing.
Time Frame: At Day 1 (survey completion visit)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group
Number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
Participants
  LE 3/1, Low parasite density | 180 | 161 | 124 | 109 | 84 | 93 | 81 | 76 | 98 | 56
  LE 3/1, Medium parasite density | 87 | 64 | 35 | 39 | 47 | 37 | 34 | 37 | 25 | 40
  LE 3/1, High parasite density | 41 | 21 | 10 | 17 | 17 | 9 | 23 | 16 | 12 | 7
  LE 3/1, Very High parasite density | 41 | 43 | 16 | 35 | 17 | 21 | 29 | 21 | 20 | 19
  LE 3/1, Negative parasite density | 561 | 337 | 284 | 410 | 1110 | 1209 | 1546 | 1525 | 1577 | 1353
  LE 3/1, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  LE 3/1, Missing |  |  |  |  | 1 |  |  |  |  |
  4-5/1, Low parasite density | 246 | 260 | 243 | 199 | 160 | 185 | 221 | 161 | 146 | 109
  4-5/1, Medium parasite density | 122 | 120 | 86 | 77 | 72 | 87 | 77 | 57 | 58 | 54
  4-5/1, High parasite density | 49 | 42 | 29 | 36 | 52 | 38 | 40 | 28 | 28 | 20
  4-5/1, Very High parasite density | 52 | 67 | 48 | 51 | 58 | 72 | 59 | 53 | 57 | 41
  4-5/1, Negative parasite density | 864 | 856 | 604 | 819 | 1439 | 1609 | 2143 | 2188 | 2299 | 2162
  4-5/1, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  4-5/1, Missing |  |  |  |  | 0 |  |  |  |  |
  GT 5/1, Low parasite density | 171 | 209 | 184 | 192 | 214 | 329 | 287 | 226 | 187 | 223
  GT 5/1, Medium parasite density | 65 | 73 | 65 | 89 | 101 | 138 | 91 | 70 | 97 | 88
  GT 5/1, High parasite density | 27 | 38 | 28 | 27 | 41 | 62 | 50 | 38 | 32 | 39
  GT 5/1, Very High parasite density | 50 | 53 | 40 | 59 | 94 | 92 | 83 | 77 | 77 | 59
  GT 5/1, Negative parasite density | 1262 | 1464 | 462 | 756 | 1488 | 1689 | 2127 | 2222 | 2099 | 2538
  GT 5/1, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  GT 5/1, Missing |  |  |  |  | 0 |  |  |  |  |
  LE 3/2, Low parasite density | 7 | 4 | 2 | 5 | 16 | 2 | 2 | 1 | 1 | 1
  LE 3/2, Medium parasite density | 2 | 0 | 1 | 1 | 8 | 0 | 0 | 1 | 1 | 0
  LE 3/2, High parasite density | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
  LE 3/2, Very High parasite density | 3 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0
  LE 3/2, Negative parasite density | 6 | 4 | 6 | 9 | 86 | 24 | 29 | 36 | 10 | 19
  LE 3/2, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  LE 3/2, Missing |  |  |  |  | 0 |  |  |  |  |
  4-5/2, Low parasite density | 8 | 14 | 20 | 8 | 12 | 10 | 12 | 16 | 8 | 10
  4-5/2, Medium parasite density | 5 | 14 | 4 | 2 | 2 | 7 | 2 | 1 | 3 | 3
  4-5/2, High parasite density | 5 | 3 | 0 | 1 | 4 | 2 | 0 | 3 | 1 | 2
  4-5/2, Very High parasite density | 4 | 3 | 1 | 0 | 6 | 1 | 0 | 1 | 5 | 0
  4-5/2, Negative parasite density | 52 | 40 | 23 | 25 | 115 | 60 | 106 | 140 | 151 | 111
  4-5/2, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  4-5/2, Missing |  |  |  |  | 0 |  |  |  |  |
  GT 5/2, Low parasite density | 8 | 21 | 20 | 7 | 12 | 28 | 25 | 8 | 15 | 23
  GT 5/2, Medium parasite density | 5 | 5 | 9 | 1 | 3 | 13 | 11 | 5 | 7 | 8
  GT 5/2, High parasite density | 4 | 7 | 3 | 1 | 4 | 4 | 0 | 4 | 2 | 4
  GT 5/2, Very High parasite density | 4 | 1 | 4 | 0 | 3 | 9 | 7 | 3 | 4 | 4
  GT 5/2, Negative parasite density | 233 | 236 | 26 | 21 | 86 | 138 | 137 | 186 | 170 | 193
  GT 5/2, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  GT 5/2, Missing |  |  |  |  | 0 |  |  |  |  |
  LE 3/3, Low parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LE 3/3, Medium parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LE 3/3, High parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LE 3/3, Very High parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LE 3/3, Negative parasite density | 3 | 0 | 0 | 0 | 18 | 0 | 0 | 0 | 0 | 0
  LE 3/3, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LE 3/3, Missing |  |  |  |  | 0 |  |  |  |  |
  4-5/3, Low parasite density | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 1 | 2 | 0
  4-5/3, Medium parasite density | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  4-5/3, High parasite density | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  4-5/3, Very High parasite density | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  4-5/3, Negative parasite density | 3 | 2 | 2 | 0 | 10 | 3 | 3 | 5 | 1 | 7
  4-5/3, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  4-5/3, Missing |  |  |  |  | 0 |  |  |  |  |
  GT 5/3, Low parasite density | 0 | 3 | 7 | 1 | 0 | 2 | 2 | 1 | 1 | 0
  GT 5/3, Medium parasite density | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
  GT 5/3, High parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  GT 5/3, Very High parasite density | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
  GT 5/3, Negative parasite density | 29 | 28 | 8 | 2 | 3 | 9 | 12 | 6 | 5 | 9
  GT 5/3, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  GT 5/3, Missing |  |  |  |  | 0 |  |  |  |  |
  4-5/GT 3, Low parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  4-5/GT 3, Medium parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  4-5/GT 3, High parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  4-5/GT 3, Very High parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  4-5/GT 3, Negative parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  4-5/GT 3, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  4-5/GT 3, Missing |  |  |  |  | 0 |  |  |  |  |
  GT 5/GT 3, Low parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  GT 5/GT 3, Medium parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  GT 5/GT 3, High parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  GT 5/GT 3, Very High parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  GT 5/GT 3, Negative parasite density | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  GT 5/GT 3, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  GT 5/GT 3, Missing |  |  |  |  | 0 |  |  |  |  |

11. Secondary Outcome: Number of Participants Experiencing Malaria Risk Categorized by Location (by Parasite Density)
Description: Participants were categorized by location as follows: situation area (rural, urban, semi-rural) and type of location (large city, small city, town, countryside). Participants were also categorized by parasite density: low (<2500 parasites/μL), medium (2500-9999/μL), high (10000-19999/μL), very high (>=20000/μL), negative, and missing.
Time Frame: At Day 1 (survey completion visit)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group
Number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
Participants
  Situation area, Rural, Low parasite density | 449 | 559 | 512 | 484 | 485 | 559 | 582 | 483 | 434 | 380
  Situation area, Rural, Medium parasite density | 210 | 252 | 195 | 203 | 226 | 250 | 202 | 169 | 183 | 178
  Situation area, Rural, High parasite density | 92 | 95 | 67 | 76 | 105 | 104 | 112 | 87 | 71 | 67
  Situation area, Rural, Very High parasite density | 109 | 150 | 102 | 133 | 169 | 166 | 170 | 155 | 159 | 116
  Situation area, Rural, Negative parasite density | 2735 | 2752 | 1231 | 1806 | 4050 | 3857 | 5498 | 6009 | 5867 | 5564
  Situation area, Rural, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Situation area, Rural, Missing |  |  |  |  | 1 |  |  |  |  |
  Situation area, Urban, Low parasite density | 158 | 6 | 3 | 2 | 6 | 3 | 9 | 3 | 6 | 7
  Situation area, Urban, Medium parasite density | 74 | 0 | 0 | 1 | 3 | 1 | 3 | 1 | 1 | 7
  Situation area, Urban, High parasite density | 32 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0
  Situation area, Urban, Very High parasite density | 41 | 1 | 0 | 1 | 3 | 1 | 4 | 1 | 3 | 1
  Situation area, Urban, Negative parasite density | 212 | 52 | 35 | 70 | 117 | 84 | 293 | 175 | 225 | 249
  Situation area, Urban, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Situation area, Urban, Missing |  |  |  |  | 0 |  |  |  |  |
  Situation area, Semi-rural, Low parasite density | 13 | 108 | 87 | 35 | 9 | 87 | 39 | 4 | 18 | 35
  Situation area, Semi-rural, Medium parasite density | 2 | 28 | 6 | 5 | 4 | 34 | 10 | 2 | 7 | 8
  Situation area, Semi-rural, High parasite density | 2 | 16 | 3 | 6 | 5 | 11 | 2 | 1 | 1 | 5
  Situation area, Semi-rural, Very High parasite density | 5 | 17 | 8 | 12 | 6 | 30 | 5 | 2 | 2 | 6
  Situation area, Semi-rural, Negative parasite density | 74 | 163 | 149 | 166 | 188 | 800 | 312 | 124 | 223 | 579
  Situation area, Semi-rural, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Situation area, Semi-rural, Missing |  |  |  |  | 0 |  |  |  |  |
  Type of location, Large city, Low parasite density | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Type of location, Large city, Medium parasite density | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Type of location, Large city, High parasite density | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Type of location, Large city, Very High parasite density | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Type of location, Large city, Negative parasite density | 10 | 2 | 0 | 3 | 0 | 1 | 6 | 0 | 19 | 4
  Type of location, Large city, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Type of location, Large city, Missing |  |  |  |  | 0 |  |  |  |  |
  Type of location, Small city, Low parasite density | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
  Type of location, Small city, Medium parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Type of location, Small city, High parasite density | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Type of location, Small city, Very High parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Type of location, Small city, Negative parasite density | 3 | 13 | 0 | 1 | 7 | 13 | 25 | 1 | 45 | 1
  Type of location, Small city, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Type of location, Small city, Missing |  |  |  |  | 0 |  |  |  |  |
  Type of location, Town, Low parasite density | 164 | 162 | 197 | 171 | 97 | 154 | 105 | 62 | 71 | 102
  Type of location, Town, Medium parasite density | 59 | 59 | 58 | 70 | 46 | 75 | 37 | 27 | 34 | 35
  Type of location, Town, High parasite density | 31 | 25 | 19 | 31 | 23 | 23 | 14 | 14 | 12 | 14
  Type of location, Town, Very High parasite density | 43 | 54 | 50 | 55 | 45 | 61 | 51 | 30 | 36 | 29
  Type of location, Town, Negative parasite density | 515 | 475 | 546 | 869 | 574 | 1067 | 1028 | 739 | 797 | 1240
  Type of location, Town, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Type of location, Town, Missing |  |  |  |  | 0 |  |  |  |  |
  Type of location, Countryside, Low parasite density | 455 | 510 | 405 | 349 | 403 | 495 | 524 | 428 | 385 | 319
  Type of location, Countryside, Medium parasite density | 226 | 220 | 143 | 139 | 187 | 210 | 178 | 145 | 156 | 158
  Type of location, Countryside, High parasite density | 95 | 84 | 52 | 51 | 87 | 91 | 100 | 75 | 63 | 58
  Type of location, Countryside, Very High parasite density | 111 | 114 | 60 | 91 | 133 | 136 | 128 | 128 | 128 | 94
  Type of location, Countryside, Negative parasite density | 2493 | 2477 | 869 | 1169 | 3774 | 3660 | 5044 | 5568 | 5454 | 5147
  Type of location, Countryside, Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Type of location, Countryside, Missing |  |  |  |  | 1 |  |  |  |  |

12. Secondary Outcome: Number of Participants Experiencing Malaria Risk Factors Categorized by House Information (by Parasite Density)
Description: Participants were categorized by house characteristics as follows: wall material (mud, brick, cement/plaster, clay, other), floor material (natural, rudimentary, vinyl/asphalt strips, parquet/polished wood, ceramic tiles, cement, carpet, clay, other), roof type (iron sheet, tiles, clay, other), window type (closed, open, no window, partially open, other), presence of nets (not present, present on all windows, present on some windows, other, missing), main drinking water source (closed, open), whether the open source was in the compound (yes, no, not available [NA]), and presence or absence of electricity. Participants were also categorized by parasite density: low (<2500 parasites/μL), medium (2500-9999/μL), high (10000-19999/μL), very high (>=20000/μL), negative, and missing.
Time Frame: At Day 1 (survey completion visit)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group
Number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
Participants
  Main house construction material of Walls: Mud, low parasite density | 417 | 500 | 218 | 257 | 217 | 322 | 298 | 231 | 202 | 161
  Main house construction material of Walls: Mud, Medium parasite density | 204 | 209 | 83 | 110 | 129 | 162 | 106 | 80 | 94 | 89
  Main house construction material of Walls: Mud, High parasite density | 97 | 81 | 38 | 48 | 59 | 75 | 55 | 44 | 38 | 32
  Main house construction material of Walls: Mud, Very High parasite density | 99 | 108 | 39 | 82 | 94 | 115 | 88 | 90 | 81 | 48
  Main house construction material of Walls: Mud, Negative parasite density | 1377 | 1375 | 643 | 1044 | 1462 | 2076 | 2306 | 2524 | 2009 | 1925
  Main house construction material of Walls: Mud, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Walls: Mud, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Walls: Brick, low parasite density | 114 | 105 | 297 | 187 | 173 | 113 | 164 | 97 | 91 | 133
  Main house construction material of Walls: Brick, Medium parasite density | 37 | 41 | 83 | 62 | 53 | 30 | 45 | 33 | 34 | 60
  Main house construction material of Walls: Brick, High parasite density | 17 | 20 | 21 | 21 | 28 | 8 | 21 | 17 | 12 | 20
  Main house construction material of Walls: Brick, very high parasite density | 21 | 31 | 36 | 46 | 32 | 23 | 40 | 21 | 23 | 31
  Main house construction material of Walls: Brick, Negative parasite density | 881 | 804 | 417 | 535 | 1841 | 1065 | 1938 | 1764 | 2055 | 2609
  Main house construction material of Walls: Brick, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Walls: Brick, missing |  |  |  |  | 1 |  |  |  |  |
  Main house construction material of Walls: Cement/Plaster, low parasite density | 57 | 46 | 37 | 54 | 66 | 134 | 136 | 135 | 84 | 86
  Main house construction material of Walls: Cement/Plaster, Medium parasite density | 25 | 16 | 14 | 31 | 22 | 66 | 51 | 50 | 35 | 29
  Main house construction material of Walls: Cement/Plaster, High parasite density | 7 | 6 | 5 | 10 | 10 | 22 | 27 | 27 | 15 | 15
  Main house construction material of Walls: Cement/Plaster, very high parasite density | 25 | 21 | 17 | 15 | 26 | 37 | 37 | 38 | 43 | 31
  Main house construction material of Walls: Cement/Plaster, Negative parasite density | 373 | 402 | 186 | 313 | 623 | 872 | 1306 | 1541 | 1163 | 1175
  Main house construction material of Walls: Cement/Plaster, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Walls: Cement/Plaster, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Walls: Cement/Paint, low parasite density | 14 | 12 | 14 | 23 | 21 | 70 | 21 | 13 | 61 | 20
  Main house construction material of Walls: Cement/Paint, Medium parasite density | 8 | 10 | 3 | 6 | 10 | 18 | 10 | 6 | 22 | 9
  Main house construction material of Walls: Cement/Paint, High parasite density | 0 | 2 | 1 | 2 | 6 | 6 | 4 | 0 | 10 | 1
  Main house construction material of Walls: Cement/Paint, very high parasite density | 6 | 1 | 4 | 3 | 16 | 18 | 8 | 6 | 13 | 5
  Main house construction material of Walls: Cement/Paint, Negative parasite density | 329 | 342 | 72 | 138 | 227 | 604 | 402 | 273 | 895 | 490
  Main house construction material of Walls: Cement/Paint, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Walls: Cement/Paint, missing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Walls: Clay, Low parasite density | 1 | 9 | 34 | 2 | 17 | 9 | 7 | 6 | 13 | 19
  Main house construction material of Walls: Clay, medium parasite density | 2 | 4 | 18 | 1 | 18 | 7 | 2 | 1 | 4 | 6
  Main house construction material of Walls: Clay, high parasite density | 0 | 2 | 6 | 1 | 7 | 2 | 6 | 1 | 0 | 4
  Main house construction material of Walls: Clay, very high parasite density | 0 | 7 | 14 | 0 | 9 | 4 | 3 | 0 | 4 | 6
  Main house construction material of Walls: Clay, negative parasite density | 6 | 40 | 96 | 10 | 167 | 70 | 104 | 84 | 127 | 111
  Main house construction material of Walls: Clay, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Walls: Clay, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Walls: Other, low parasite density | 17 | 1 | 2 | 1 | 6 | 1 | 4 | 8 | 7 | 3
  Main house construction material of Walls: Other, medium parasite density | 10 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 2 | 0
  Main house construction material of Walls: Other, high parasite density | 5 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
  Main house construction material of Walls: Other, very high parasite density | 4 | 0 | 0 | 0 | 1 | 0 | 3 | 3 | 0 | 2
  Main house construction material of Walls: Other, negative parasite density | 55 | 4 | 1 | 2 | 35 | 54 | 47 | 122 | 66 | 82
  Main house construction material: Walls: Other, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material: Walls: Other, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Floor: Natural floor, low parasite density | 248 | 325 | 223 | 204 | 217 | 263 | 228 | 171 | 167 | 171
  Main house construction material of Floor: Natural floor, medium parasite density | 133 | 140 | 85 | 76 | 124 | 131 | 88 | 69 | 85 | 85
  Main house construction material of Floor: Natural floor, high parasite density | 63 | 49 | 27 | 32 | 54 | 55 | 46 | 24 | 28 | 28
  Main house construction material of Floor: Natural floor, very high parasite density | 61 | 84 | 37 | 57 | 84 | 83 | 69 | 74 | 66 | 45
  Main house construction material of Floor: Natural floor, negative parasite density | 1173 | 1384 | 506 | 652 | 1615 | 1730 | 1963 | 1844 | 2063 | 1851
  Main house construction material of Floor: Natural floor, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Floor: Natural floor, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Floor: Rudimentary floor, low parasite density: number analyzed (Participants) | 4208 | 0 | 2399 | 0 | 0 | 0 | 7241 | 7217 | 0 | 7202
  Main house construction material of Floor: Rudimentary floor, low parasite density | 0 |  | 3 |  |  |  | 0 | 1 |  | 0
  Main house construction material of Floor: Rudimentary floor, medium parasite density: number analyzed (Participants) | 4208 | 0 | 2399 | 0 | 0 | 0 | 7241 | 7217 | 0 | 7202
  Main house construction material of Floor: Rudimentary floor, medium parasite density | 0 |  | 0 |  |  |  | 0 | 0 |  | 0
  Main house construction material of Floor: Rudimentary floor, high parasite density: number analyzed (Participants) | 4208 | 0 | 2399 | 0 | 0 | 0 | 7241 | 0 | 0 | 7202
  Main house construction material of Floor: Rudimentary floor, high parasite density | 0 |  | 1 |  |  |  | 0 | 0 |  | 0
  Main house construction material of Floor: Rudimentary floor, very high parasite density: number analyzed (Participants) | 4208 | 0 | 2399 | 0 | 0 | 0 | 7241 | 7217 | 0 | 7202
  Main house construction material of Floor: Rudimentary floor, very high parasite density | 0 |  | 3 |  |  |  | 0 | 3 |  | 0
  Main house construction material of Floor: Rudimentary floor, negative parasite density: number analyzed (Participants) | 4208 | 0 | 2399 | 0 | 0 | 0 | 7241 | 7217 | 0 | 7202
  Main house construction material of Floor: Rudimentary floor, negative parasite density | 1 |  | 13 |  |  |  | 1 | 122 |  | 1
  Main house construction material of Floor: Rudimentary floor, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Floor: Vinyl or asphalt strips, low parasite density: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7202
  Main house construction material of Floor: Vinyl or asphalt strips, low parasite density |  |  |  |  |  |  |  |  |  | 0
  Main house construction material of Floor: Vinyl or asphalt strips, medium parasite density: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7202
  Main house construction material of Floor: Vinyl or asphalt strips, medium parasite density |  |  |  |  |  |  |  |  |  | 0
  Main house construction material of Floor: Vinyl or asphalt strips, high parasite density: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7202
  Main house construction material of Floor: Vinyl or asphalt strips, high parasite density |  |  |  |  |  |  |  |  |  | 0
  Main house construction material of Floor: Vinyl or asphalt strips, very high parasite density: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7202
  Main house construction material of Floor: Vinyl or asphalt strips, very high parasite density |  |  |  |  |  |  |  |  |  | 0
  Main house construction material of Floor: Vinyl or asphalt strips, negative parasite density: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7202
  Main house construction material of Floor: Vinyl or asphalt strips, negative parasite density |  |  |  |  |  |  |  |  |  | 1
  Main house construction material of Floor: Vinyl or asphalt strips, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Floor: Parquet/ polished wood, low parasite density: number analyzed (Participants) | 0 | 4199 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Floor: Parquet/ polished wood, low parasite density |  | 0 |  |  |  |  |  |  |  |
  Main house construction material of Floor: Parquet/ polished wood, medium parasite density: number analyzed (Participants) | 0 | 4199 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Floor: Parquet/ polished wood, medium parasite density |  | 0 |  |  |  |  |  |  |  |
  Main house construction material of Floor: Parquet/ polished wood, high parasite density: number analyzed (Participants) | 0 | 4199 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Floor: Parquet/ polished wood, high parasite density |  | 0 |  |  |  |  |  |  |  |
  Main house construction material of Floor: Parquet/ polished wood, very high parasite density: number analyzed (Participants) | 0 | 4199 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Floor: Parquet/ polished wood, very high parasite density |  | 0 |  |  |  |  |  |  |  |
  Main house construction material of Floor: Parquet/ polished wood, negative parasite density: number analyzed (Participants) | 0 | 4199 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Floor: Parquet/ polished wood, negative parasite density |  | 1 |  |  |  |  |  |  |  |
  Main house construction material of Floor: Ceramic tiles, low parasite density | 1 | 0 | 6 | 1 | 3 | 7 | 5 | 4 | 10 | 5
  Main house construction material of Floor: Ceramic tiles, medium parasite density | 1 | 0 | 0 | 3 | 0 | 6 | 1 | 2 | 5 | 4
  Main house construction material of Floor: Ceramic tiles, high parasite density | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1
  Main house construction material of Floor: Ceramic tiles, very high parasite density | 0 | 1 | 2 | 1 | 1 | 3 | 3 | 6 | 9 | 2
  Main house construction material of Floor: Ceramic tiles, negative parasite density | 60 | 70 | 13 | 10 | 41 | 89 | 104 | 169 | 217 | 192
  Main house construction material of Floor: Ceramic tiles, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Floor: Ceramic tiles, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Floor: Cement, low parasite density: number analyzed (Participants) | 4208 | 0 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
  Main house construction material of Floor: Cement, low parasite density | 336 |  | 327 | 305 | 209 | 290 | 304 | 264 | 172 | 193
  Main house construction material of Floor: Cement, medium parasite density: number analyzed (Participants) | 4208 | 0 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
  Main house construction material of Floor: Cement, medium parasite density | 136 |  | 101 | 124 | 80 | 114 | 98 | 80 | 70 | 77
  Main house construction material of Floor: Cement, high parasite density: number analyzed (Participants) | 4208 | 0 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
  Main house construction material of Floor: Cement, high parasite density | 54 |  | 37 | 49 | 37 | 43 | 46 | 56 | 33 | 32
  Main house construction material of Floor: Cement, very high parasite density: number analyzed (Participants) | 4208 | 0 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
  Main house construction material of Floor: Cement, very high parasite density | 84 |  | 51 | 87 | 78 | 83 | 74 | 62 | 67 | 56
  Main house construction material of Floor: Cement, negative parasite density: number analyzed (Participants) | 4208 | 0 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
  Main house construction material of Floor: Cement, negative parasite density | 1686 |  | 773 | 1313 | 1790 | 2143 | 2855 | 3075 | 2527 | 2900
  Main house construction material of Floor: Cement, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Floor: Cement, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Floor: Carpet, low parasite density | 3 | 0 | 1 | 6 | 2 | 39 | 4 | 1 | 47 | 12
  Main house construction material of Floor: Carpet, medium parasite density | 1 | 0 | 0 | 2 | 0 | 13 | 0 | 1 | 14 | 1
  Main house construction material of Floor: Carpet, high parasite density | 1 | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 6 | 2
  Main house construction material of Floor: Carpet, very high parasite density | 1 | 0 | 0 | 0 | 0 | 10 | 4 | 0 | 8 | 2
  Main house construction material of Floor: Carpet, negative parasite density | 87 | 28 | 2 | 32 | 19 | 358 | 87 | 48 | 630 | 343
  Main house construction material of Floor: Carpet, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Floor: Carpet, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Floor: Clay, low parasite density | 32 | 30 | 42 | 5 | 69 | 43 | 89 | 43 | 52 | 41
  Main house construction material of Floor: Clay, medium parasite density | 15 | 11 | 15 | 3 | 29 | 18 | 27 | 20 | 16 | 26
  Main house construction material of Floor: Clay, high parasite density | 7 | 3 | 6 | 1 | 17 | 8 | 20 | 6 | 8 | 8
  Main house construction material of Floor: Clay, very high parasite density | 9 | 4 | 17 | 11 | 15 | 15 | 29 | 15 | 14 | 18
  Main house construction material of Floor: Clay, negative parasite density | 14 | 6 | 108 | 13 | 886 | 362 | 1088 | 1124 | 847 | 1103
  Main house construction material of Floor: Clay, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Floor: Clay, missing |  |  |  |  | 1 |  |  |  |  |
  Main house construction material of Floor: Other, low parasite density: number analyzed (Participants) | 0 | 0 | 0 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
  Main house construction material of Floor: Other, low parasite density |  |  |  | 0 | 0 | 7 | 0 | 6 | 10 | 0
  Main house construction material of Floor: Other, medium parasite density: number analyzed (Participants) | 0 | 0 | 0 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
  Main house construction material of Floor: Other, medium parasite density |  |  |  | 1 | 0 | 3 | 1 | 0 | 1 | 0
  Main house construction material of Floor: Other, high parasite density: number analyzed (Participants) | 0 | 0 | 0 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
  Main house construction material of Floor: Other, high parasite density |  |  |  | 0 | 1 | 3 | 0 | 3 | 0 | 1
  Main house construction material of Floor: Other, very high parasite density: number analyzed (Participants) | 0 | 0 | 0 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
  Main house construction material of Floor: Other, very high parasite density |  |  |  | 0 | 0 | 3 | 0 | 1 | 0 | 0
  Main house construction material of Floor: Other, negative parasite density: number analyzed (Participants) | 0 | 0 | 0 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
  Main house construction material of Floor: Other, negative parasite density |  |  |  | 21 | 3 | 59 | 5 | 46 | 31 | 1
  Main house construction material of Floor: Other, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Floor: Other, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Roof: Grass/Palm, low parasite density | 128 | 89 | 71 | 50 | 115 | 90 | 116 | 67 | 74 | 57
  Main house construction material of Roof: Grass/Palm, medium parasite density | 58 | 42 | 23 | 21 | 52 | 32 | 31 | 26 | 20 | 35
  Main house construction material of Roof: Grass/Palm, high parasite density | 29 | 12 | 13 | 5 | 22 | 10 | 19 | 16 | 10 | 10
  Main house construction material of Roof: Grass/Palm, very high parasite density | 20 | 22 | 14 | 10 | 30 | 25 | 26 | 18 | 18 | 20
  Main house construction material of Roof: Grass/Palm, negative parasite density | 784 | 703 | 197 | 140 | 1187 | 807 | 1278 | 1301 | 1165 | 1198
  Main house construction material of Roof: Grass/Palm, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Roof: Grass/Palm, missing |  |  |  |  | 1 |  |  |  |  |
  Main house construction material of Roof: Iron sheet, low parasite density | 386 | 462 | 445 | 418 | 371 | 540 | 486 | 407 | 365 | 353
  Main house construction material of Roof: Iron sheet, medium parasite density | 170 | 201 | 159 | 172 | 178 | 236 | 175 | 138 | 161 | 154
  Main house construction material of Roof: Iron sheet, high parasite density | 72 | 84 | 57 | 70 | 86 | 99 | 88 | 68 | 63 | 55
  Main house construction material of Roof: Iron sheet, very high parasite density | 107 | 129 | 90 | 115 | 147 | 163 | 149 | 135 | 136 | 100
  Main house construction material of Roof: Iron sheet, negative parasite density | 2111 | 2205 | 1144 | 1729 | 3056 | 3728 | 4636 | 4824 | 5026 | 5081
  Main house construction material of Roof: Iron sheet, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Roof: Iron sheet, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Roof: Tiles, low parasite density: number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 0 | 7202
  Main house construction material of Roof: Tiles, low parasite density | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  Main house construction material of Roof: Tiles, medium parasite density: number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 0 | 7202
  Main house construction material of Roof: Tiles, medium parasite density | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 |  | 0
  Main house construction material of Roof: Tiles, high parasite density: number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 0 | 7202
  Main house construction material of Roof: Tiles, high parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  Main house construction material of Roof: Tiles, very high parasite density: number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 0 | 7202
  Main house construction material of Roof: Tiles, very high parasite density | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  Main house construction material of Roof: Tiles, negative parasite density: number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 0 | 7202
  Main house construction material of Roof: Tiles, negative parasite density | 18 | 18 | 3 | 2 | 4 | 3 | 3 | 5 |  | 3
  Main house construction material of Roof: Tiles, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Roof: Tiles, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Roof: Clay, low parasite density | 97 | 120 | 86 | 42 | 13 | 2 | 0 | 5 | 7 | 5
  Main house construction material of Roof: Clay, medium parasite density | 55 | 36 | 17 | 9 | 3 | 2 | 0 | 5 | 3 | 2
  Main house construction material of Roof: Clay, high parasite density | 25 | 15 | 1 | 5 | 2 | 0 | 2 | 1 | 2 | 5
  Main house construction material of Roof: Clay, very high parasite density | 27 | 17 | 6 | 9 | 1 | 0 | 1 | 1 | 2 | 1
  Main house construction material of Roof: Clay, negative parasite density | 61 | 39 | 71 | 80 | 100 | 17 | 8 | 47 | 47 | 65
  Main house construction material of Roof: Clay, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Roof: Clay, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Roof: Other, low parasite density: number analyzed (Participants) | 4208 | 4199 | 0 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
  Main house construction material of Roof: Other, low parasite density | 8 | 0 |  | 11 | 1 | 17 | 28 | 11 | 12 | 7
  Main house construction material of Roof: Other, medium parasite density: number analyzed (Participants) | 4208 | 4199 | 0 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
  Main house construction material of Roof: Other, medium parasite density | 3 | 1 |  | 7 | 0 | 15 | 9 | 3 | 7 | 2
  Main house construction material of Roof: Other, high parasite density: number analyzed (Participants) | 4208 | 4199 | 0 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
  Main house construction material of Roof: Other, high parasite density | 0 | 0 |  | 2 | 0 | 6 | 5 | 4 | 0 | 2
  Main house construction material of Roof: Other, very high parasite density: number analyzed (Participants) | 4208 | 4199 | 0 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
  Main house construction material of Roof: Other, very high parasite density | 1 | 0 |  | 12 | 0 | 9 | 3 | 4 | 8 | 2
  Main house construction material of Roof: Other, negative parasite density: number analyzed (Participants) | 4208 | 4199 | 0 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
  Main house construction material of Roof: Other, negative parasite density | 47 | 2 |  | 91 | 8 | 186 | 178 | 131 | 77 | 45
  Main house construction material of Roof: Other, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Roof: Other, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Windows/eaves: Closed, low parasite density | 236 | 236 | 286 | 253 | 115 | 179 | 131 | 123 | 123 | 130
  Main house construction material of Windows/eaves: Closed, medium parasite density | 115 | 103 | 79 | 104 | 46 | 66 | 51 | 46 | 53 | 59
  Main house construction material of Windows/eaves: Closed, high parasite density | 44 | 45 | 32 | 34 | 24 | 32 | 33 | 11 | 25 | 17
  Main house construction material of Windows/eaves: Closed, very high parasite density | 44 | 48 | 35 | 69 | 38 | 56 | 30 | 32 | 33 | 28
  Main house construction material of Windows/eaves: Closed, negative parasite density | 677 | 487 | 587 | 911 | 1023 | 1368 | 1251 | 1494 | 1964 | 2109
  Main house construction material of Windows/eaves: Closed, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Windows/eaves: Closed, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Windows/eaves: No Windows, low parasite density | 139 | 111 | 40 | 60 | 112 | 149 | 122 | 87 | 109 | 89
  Main house construction material of Windows/eaves: No Windows, medium parasite density | 67 | 45 | 25 | 23 | 75 | 86 | 61 | 40 | 50 | 58
  Main house construction material of Windows/eaves: No Windows, high parasite density | 36 | 17 | 7 | 9 | 36 | 36 | 34 | 24 | 20 | 25
  Main house construction material of Windows/eaves: No Windows, very high parasite density | 29 | 35 | 15 | 13 | 64 | 47 | 53 | 51 | 43 | 28
  Main house construction material of Windows/eaves: No Windows, negative parasite density | 942 | 821 | 124 | 143 | 660 | 911 | 1063 | 987 | 956 | 944
  Main house construction material of Windows/eaves: No Windows, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Windows/eaves: No Windows, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Windows/eaves: Open, low parasite density | 209 | 215 | 170 | 151 | 197 | 182 | 173 | 197 | 150 | 107
  Main house construction material of Windows/eaves: Open, medium parasite density | 83 | 84 | 52 | 58 | 87 | 73 | 37 | 66 | 62 | 30
  Main house construction material of Windows/eaves: Open, high parasite density | 37 | 32 | 10 | 31 | 39 | 19 | 25 | 38 | 15 | 13
  Main house construction material of Windows/eaves: Open, very high parasite density | 67 | 54 | 30 | 44 | 58 | 42 | 47 | 63 | 51 | 27
  Main house construction material of Windows/eaves: Open, negative parasite density | 1189 | 1050 | 353 | 662 | 1902 | 1352 | 1961 | 2723 | 2087 | 1819
  Main house construction material of Windows/eaves: Open missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Windows/eaves: Open missing |  |  |  |  | 1 |  |  |  |  |
  Main house construction material of Windows/eaves: Partially open, low parasite density | 35 | 111 | 106 | 57 | 76 | 139 | 204 | 83 | 76 | 96
  Main house construction material of Windows/eaves: Partially open, medium parasite density | 21 | 48 | 45 | 24 | 25 | 60 | 66 | 30 | 26 | 46
  Main house construction material of Windows/eaves: Partially open, high parasite density | 9 | 17 | 22 | 8 | 11 | 28 | 22 | 16 | 15 | 17
  Main house construction material of Windows/eaves: Partially open, very high parasite density | 15 | 31 | 30 | 20 | 18 | 52 | 49 | 12 | 37 | 40
  Main house construction material of Windows/eaves: Partially open, negative parasite density | 206 | 571 | 351 | 326 | 769 | 1108 | 1828 | 1104 | 1308 | 1518
  Main house construction material of Windows/eaves: Partially open, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Windows/eaves: Partially open, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Windows/eaves: Other, low parasite density: number analyzed (Participants) | 4208 | 4199 | 0 | 0 | 5377 | 5987 | 0 | 0 | 0 | 7202
  Main house construction material of Windows/eaves: Other, low parasite density | 1 | 0 |  |  | 0 | 0 |  |  |  | 0
  Main house construction material of Windows/eaves: Other, medium parasite density: number analyzed (Participants) | 4208 | 4199 | 0 | 0 | 5377 | 5987 | 0 | 0 | 0 | 7202
  Main house construction material of Windows/eaves: Other, medium parasite density | 0 | 0 |  |  | 0 | 0 |  |  |  | 0
  Main house construction material of Windows/eaves: Other, high parasite density: number analyzed (Participants) | 4208 | 4199 | 0 | 0 | 5377 | 5987 | 0 | 0 | 0 | 7202
  Main house construction material of Windows/eaves: Other, high parasite density | 0 | 0 |  |  | 0 | 0 |  |  |  | 0
  Main house construction material of Windows/eaves: Other, very high parasite density: number analyzed (Participants) | 4208 | 4199 | 0 | 0 | 5377 | 5987 | 0 | 0 | 0 | 7202
  Main house construction material of Windows/eaves: Other, very high parasite density | 0 | 0 |  |  | 0 | 0 |  |  |  | 0
  Main house construction material of Windows/eaves: Other, negative parasite density: number analyzed (Participants) | 4208 | 4199 | 0 | 0 | 5377 | 5987 | 0 | 0 | 0 | 7202
  Main house construction material of Windows/eaves: Other, negative parasite density | 7 | 38 |  |  | 1 | 2 |  |  |  | 2
  Main house construction material of Windows/eaves: Other, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Windows/eaves: Other, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Nets: Nets not present, low parasite density | 505 | 506 | 499 | 393 | 269 | 340 | 366 | 290 | 244 | 230
  Main house construction material of Nets: Nets not present, medium parasite density | 231 | 216 | 152 | 160 | 114 | 148 | 118 | 103 | 107 | 103
  Main house construction material of Nets: Nets not present, high parasite density | 101 | 85 | 56 | 59 | 55 | 59 | 62 | 46 | 40 | 32
  Main house construction material of Nets: Nets not present, very high parasite density | 117 | 114 | 77 | 117 | 83 | 91 | 99 | 89 | 97 | 66
  Main house construction material of Nets: Nets not present, negative parasite density | 2313 | 1550 | 1100 | 1407 | 2765 | 2486 | 3636 | 3724 | 3728 | 3730
  Main house construction material of Nets: Nets not present, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Nets: Nets not present, missing |  |  |  |  | 1 |  |  |  |  |
  Main house construction material of Nets: Nets present on all windows, low parasite density | 32 | 48 | 58 | 60 | 101 | 147 | 129 | 104 | 100 | 84
  Main house construction material of Nets: Nets present on all windows, medium parasite density | 19 | 18 | 23 | 22 | 40 | 44 | 32 | 28 | 33 | 25
  Main house construction material of Nets: Nets present on all windows, high parasite density | 5 | 7 | 7 | 12 | 17 | 20 | 17 | 17 | 14 | 9
  Main house construction material of Nets: Nets present on all windows, very high parasite density | 16 | 17 | 16 | 15 | 29 | 50 | 26 | 18 | 23 | 22
  Main house construction material of Nets: Nets present on all windows, negative parasite density | 322 | 411 | 180 | 434 | 773 | 1207 | 1290 | 1462 | 1496 | 1422
  Main house construction material of Nets: Nets present on all windows, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Nets: Nets present on all windows, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Nets: Nets present on some windows, low parasite density | 12 | 7 | 5 | 8 | 12 | 13 | 11 | 8 | 4 | 17
  Main house construction material of Nets: Nets present on some windows, medium parasite density | 6 | 0 | 1 | 4 | 3 | 7 | 4 | 1 | 1 | 2
  Main house construction material of Nets: Nets present on some windows, high parasite density | 2 | 2 | 1 | 2 | 1 | 0 | 1 | 2 | 1 | 5
  Main house construction material of Nets: Nets present on some windows, very high parasite density | 5 | 1 | 1 | 1 | 1 | 9 | 1 | 0 | 0 | 5
  Main house construction material of Nets: Nets present on some windows, negative parasite density | 99 | 88 | 11 | 57 | 130 | 135 | 103 | 124 | 118 | 216
  Main house construction material of Nets: Nets present on some windows, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Nets: Nets present on some windows, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Nets: Other, low parasite density | 71 | 112 | 40 | 60 | 94 | 149 | 124 | 88 | 110 | 91
  Main house construction material of Nets: Other, medium parasite density | 30 | 46 | 25 | 23 | 66 | 86 | 61 | 1 | 50 | 63
  Main house construction material of Nets: Other, high parasite density | 18 | 17 | 7 | 9 | 23 | 36 | 34 | 2 | 20 | 26
  Main house construction material of Nets: Other, very high parasite density | 17 | 36 | 16 | 13 | 47 | 47 | 53 | 0 | 44 | 30
  Main house construction material of Nets: Other, negative parasite density | 287 | 918 | 124 | 144 | 557 | 913 | 1074 | 124 | 973 | 1024
  Main house construction material of Nets: Other, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Nets: Other, missing |  |  |  |  | 0 |  |  |  |  |
  Main house construction material of Nets: Missing, low parasite density: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Nets: Missing, low parasite density |  |  |  |  | 24 |  |  |  |  |
  Main house construction material of Nets: Missing, medium parasite density: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Nets: Missing, medium parasite density |  |  |  |  | 10 |  |  |  |  |
  Main house construction material of Nets: Missing, high parasite density: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Nets: Missing, high parasite density |  |  |  |  | 14 |  |  |  |  |
  Main house construction material of Nets: Missing, very high parasite density: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Nets: Missing, very high parasite density |  |  |  |  | 18 |  |  |  |  |
  Main house construction material of Nets: Missing, negative parasite density: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Nets: Missing, negative parasite density |  |  |  |  | 130 |  |  |  |  |
  Main house construction material of Nets: Missing, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main house construction material of Nets: Missing, missing |  |  |  |  | 0 |  |  |  |  |
  Main source of the drinking water: Closed water source, low parasite density | 388 | 357 | 377 | 334 | 366 | 438 | 461 | 340 | 322 | 280
  Main source of the drinking water: Closed water source, medium parasite density | 172 | 145 | 116 | 139 | 144 | 160 | 127 | 112 | 129 | 128
  Main source of the drinking water: Closed water source, high parasite density | 67 | 66 | 52 | 53 | 63 | 68 | 81 | 57 | 48 | 45
  Main source of the drinking water: Closed water source, very high parasite density | 94 | 91 | 72 | 91 | 103 | 126 | 112 | 85 | 103 | 78
  Main source of the drinking water: Closed water source, negative parasite density | 2070 | 1948 | 1002 | 1491 | 3455 | 3546 | 4730 | 4958 | 4984 | 4973
  Main source of the drinking water: Closed water source, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main source of the drinking water: Closed water source, missing |  |  |  |  | 1 |  |  |  |  |
  Main source of the drinking water: Open water source, low parasite density | 232 | 316 | 225 | 187 | 134 | 211 | 169 | 150 | 136 | 142
  Main source of the drinking water: Open water source, medium parasite density | 114 | 135 | 85 | 70 | 89 | 125 | 88 | 60 | 62 | 65
  Main source of the drinking water: Open water source, high parasite density | 59 | 45 | 19 | 29 | 47 | 47 | 33 | 32 | 27 | 27
  Main source of the drinking water: Open water source, very high parasite density | 61 | 77 | 38 | 55 | 75 | 71 | 67 | 73 | 61 | 45
  Main source of the drinking water: Open water source, negative parasite density | 951 | 1019 | 413 | 551 | 900 | 1195 | 1373 | 1350 | 1331 | 1419
  Main source of the drinking water: Open water source, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Main source of the drinking water: Open water source, missing |  |  |  |  | 0 |  |  |  |  |
  The open source is in compound: Yes, low parasite density | 64 | 98 | 57 | 17 | 27 | 34 | 29 | 9 | 26 | 32
  The open source is in compound: Yes, medium parasite density | 21 | 34 | 10 | 8 | 7 | 25 | 11 | 5 | 13 | 12
  The open source is in compound: Yes, high parasite density | 12 | 10 | 2 | 4 | 7 | 7 | 0 | 1 | 3 | 3
  The open source is in compound: Yes, very high parasite density | 17 | 14 | 7 | 9 | 9 | 16 | 14 | 5 | 9 | 8
  The open source is in compound: Yes, negative parasite density | 253 | 250 | 72 | 93 | 133 | 175 | 212 | 149 | 251 | 272
  The open source is in compound: Yes, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  The open source is in compound: Yes, missing |  |  |  |  | 0 |  |  |  |  |
  The open source is in compound: No, low parasite density | 168 | 218 | 168 | 170 | 107 | 177 | 140 | 141 | 110 | 110
  The open source is in compound: No, medium parasite density | 93 | 101 | 75 | 62 | 82 | 100 | 77 | 55 | 49 | 53
  The open source is in compound: No, high parasite density | 47 | 35 | 17 | 25 | 40 | 40 | 33 | 31 | 24 | 24
  The open source is in compound: No, very high parasite density | 44 | 63 | 31 | 46 | 66 | 55 | 53 | 68 | 52 | 37
  The open source is in compound: No, negative parasite density | 698 | 769 | 341 | 458 | 767 | 1020 | 1161 | 1201 | 1080 | 1147
  The open source is in compound: No, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  The open source is in compound: No, missing |  |  |  |  | 0 |  |  |  |  |
  The open source is in compound: NA, low parasite density | 388 | 357 | 377 | 334 | 366 | 438 | 461 | 340 | 322 | 280
  The open source is in compound: NA, medium parasite density | 172 | 145 | 116 | 139 | 144 | 160 | 127 | 112 | 129 | 128
  The open source is in compound: NA, high parasite density | 67 | 66 | 52 | 53 | 63 | 68 | 81 | 57 | 48 | 45
  The open source is in compound: NA, very high parasite density | 94 | 91 | 72 | 91 | 103 | 126 | 112 | 85 | 103 | 78
  The open source is in compound: NA, negative parasite density | 2070 | 1948 | 1002 | 1491 | 3455 | 3546 | 4730 | 4958 | 4984 | 4973
  The open source is in compound: NA, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  The open source is in compound: NA, missing |  |  |  |  | 1 |  |  |  |  |
  Number of participants in houses with the presence of electricity, low parasite density | 98 | 210 | 230 | 232 | 163 | 184 | 180 | 134 | 126 | 108
  Number of participants in houses with the presence of electricity, medium parasite density | 45 | 80 | 51 | 88 | 83 | 38 | 40 | 36 | 49 | 39
  Number of participants in houses with the presence of electricity, high parasite density | 8 | 39 | 11 | 35 | 38 | 26 | 20 | 19 | 15 | 15
  Number of participants in houses with the presence of electricity, very high parasite density | 30 | 40 | 26 | 48 | 75 | 56 | 41 | 28 | 41 | 35
  Number of participants in houses with the presence of electricity, negative parasite density | 637 | 631 | 446 | 946 | 1481 | 1574 | 1722 | 1968 | 2112 | 2175
  Number of participants in houses with the presence of electricity, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Number of participants in houses with the presence of electricity, missing |  |  |  |  | 0 |  |  |  |  |
  Number of participants in houses with no presence of electricity, low parasite density | 522 | 463 | 372 | 289 | 337 | 465 | 450 | 356 | 332 | 314
  Number of participants in houses with no presence of electricity, medium parasite density | 241 | 200 | 150 | 121 | 150 | 247 | 175 | 136 | 142 | 154
  Number of participants in houses with no presence of electricity, high parasite density | 118 | 72 | 60 | 47 | 72 | 89 | 94 | 70 | 60 | 57
  Number of participants in houses with no presence of electricity, very high parasite density | 125 | 128 | 84 | 98 | 103 | 141 | 138 | 130 | 123 | 88
  Number of participants in houses with no presence of electricity, negative parasite density | 2384 | 2336 | 969 | 1096 | 2975 | 3167 | 4381 | 4340 | 4203 | 4217
  Number of participants in houses with no presence of electricity, missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 0 | 0
  Number of participants in houses with no presence of electricity, missing |  |  |  |  | 1 |  |  |  |  |

13. Primary Outcome: Number of Participants Infected With P. Falciparum by Joint Technical Expert Group (JTEG) Age Group
Description: The number of participants was summarized by the JTEG age group (0.5-4Y and 5-9Y) by center number/ country [BF, SN, TZ, KE, GH, MA]/ city. UNEXP sites are the ones in which the RTS,S vaccine was not planned to be implemented during the course of the study however, vaccinated participants could still have been randomly selected in this population if vaccination happened in an EXP site, due to cross-site migration. The infection was identified using a blood smear slide and determined using microscopy.
Time Frame: At Day 1 (survey completion visit)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group
Number analyzed (Participants) | 404 | 401 | 401 | 403 | 405 | 402 | 415 | 412 | 403 | 408
Participants
  0.5-4Y, 207078_BF_Nouna: number analyzed (Participants) | 404 | 400 | 400 | 401 | 0 | 0 | 0 | 0 | 0 | 0
  0.5-4Y, 207078_BF_Nouna | 249 | 321 | 198 | 135 |  |  |  |  |  |
  0.5-4Y, 207079_BF_Sapone: number analyzed (Participants) | 403 | 399 | 401 | 399 | 0 | 0 | 0 | 0 | 0 | 0
  0.5-4Y, 207079_BF_Sapone | 162 | 182 | 75 | 94 |  |  |  |  |  |
  0.5-4Y, 207080_SN_Niakhar: number analyzed (Participants) | 398 | 397 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  0.5-4Y, 207080_SN_Niakhar | 6 | 1 |  |  |  |  |  |  |  |
  0.5-4Y, 207081_TZ_Korogwe: number analyzed (Participants) | 401 | 400 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  0.5-4Y, 207081_TZ_Korogwe | 29 | 6 |  |  |  |  |  |  |  |
  0.5-4Y, 207082_KE_Kombewa: number analyzed (Participants) | 402 | 401 | 401 | 403 | 402 | 399 | 400 | 402 | 401 | 397
  0.5-4Y, 207082_KE_Kombewa | 100 | 108 | 119 | 132 | 109 | 111 | 76 | 68 | 64 | 51
  0.5-4Y, 207083_GH_Kintampo: number analyzed (Participants) | 400 | 400 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  0.5-4Y, 207083_GH_Kintampo | 99 | 109 |  |  |  |  |  |  |  |
  0 .5-4Y, 207083_GH_Kintampo_EXP: number analyzed (Participants) | 0 | 0 | 401 | 398 | 401 | 402 | 400 | 398 | 400 | 400
  0 .5-4Y, 207083_GH_Kintampo_EXP |  |  | 117 | 103 | 40 | 53 | 45 | 25 | 24 | 23
  0.5-4Y, 207083_GH_Kintampo_UNEXP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 401 | 399 | 403 | 399 | 399
  0.5-4Y, 207083_GH_Kintampo_UNEXP |  |  |  |  | 0 | 81 | 66 | 58 | 42 | 33
  0.5-4Y, 207084_SN_Keur Soce: number analyzed (Participants) | 400 | 397 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  0.5-4Y, 207084_SN_Keur Soce | 2 | 4 |  |  |  |  |  |  |  |
  0 .5-4Y, 228607_GH_Navrongo_EXP: number analyzed (Participants) | 0 | 0 | 0 | 403 | 401 | 400 | 398 | 399 | 400 | 400
  0 .5-4Y, 228607_GH_Navrongo_EXP |  |  |  | 31 | 40 | 32 | 19 | 14 | 25 | 22
  0.5-4Y, 228607_GH_Navrongo_UNEXP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 400 | 401 | 399 | 399 | 407
  0.5-4Y, 228607_GH_Navrongo_UNEXP |  |  |  |  |  | 26 | 28 | 27 | 28 | 36
  0 .5-4Y, 233149_MA_Mangochi: number analyzed (Participants) | 0 | 0 | 0 | 0 | 399 | 398 | 402 | 389 | 399 | 400
  0 .5-4Y, 233149_MA_Mangochi |  |  |  |  | 51 | 39 | 27 | 34 | 24 | 28
  0 .5-4Y, 233149_MA_Monkey Bay: number analyzed (Participants) | 0 | 0 | 0 | 0 | 395 | 400 | 399 | 406 | 397 | 403
  0 .5-4Y, 233149_MA_Monkey Bay |  |  |  |  | 27 | 8 | 18 | 15 | 19 | 22
  0 .5-4Y, 233150_MA_Chikwawa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 391 | 0 | 415 | 398 | 399 | 397
  0 .5-4Y, 233150_MA_Chikwawa |  |  |  |  | 33 | 0 | 43 | 10 | 7 | 12
  0 .5-4Y, 233150_MA_St Monfort: number analyzed (Participants) | 0 | 0 | 0 | 0 | 389 | 0 | 414 | 402 | 399 | 401
  0 .5-4Y, 233150_MA_St Monfort |  |  |  |  | 17 |  | 27 | 5 | 0 | 2
  0 .5-4Y, 235578_KE_Bondo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 405 | 390 | 405 | 405 | 403 | 400
  0 .5-4Y, 235578_KE_Bondo |  |  |  |  | 94 | 99 | 74 | 63 | 55 | 44
  0 .5-4Y, 235578_KE_Gem: number analyzed (Participants) | 0 | 0 | 0 | 0 | 402 | 393 | 402 | 405 | 398 | 402
  0 .5-4Y, 235578_KE_Gem |  |  |  |  | 80 | 64 | 48 | 55 | 48 | 43
  0.5-4Y, 235579_KE_Nyando: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 397 | 395 | 412 | 403 | 408
  0.5-4Y, 235579_KE_Nyando |  |  |  |  | 0 | 83 | 48 | 41 | 43 | 39
  5-9Y, 207078_BF_Nouna: number analyzed (Participants) | 202 | 200 | 200 | 199 | 0 | 0 | 0 | 0 | 0 | 0
  5-9Y, 207078_BF_Nouna | 154 | 167 | 154 | 122 |  |  |  |  |  |
  5-9Y, 207079_BF_Sapone: number analyzed (Participants) | 201 | 200 | 199 | 201 | 0 | 0 | 0 | 0 | 0 | 0
  5-9Y, 207079_BF_Sapone | 137 | 134 | 119 | 110 |  |  |  |  |  |
  5-9Y, 207080_SN_Niakhar: number analyzed (Participants) | 200 | 204 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  5-9Y, 207080_SN_Niakhar | 3 | 2 |  |  |  |  |  |  |  |
  5-9Y, 207081_TZ_Korogwe: number analyzed (Participants) | 200 | 200 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  5-9Y, 207081_TZ_Korogwe | 34 | 12 |  |  |  |  |  |  |  |
  5-9Y, 207082_KE_Kombewa: number analyzed (Participants) | 197 | 198 | 198 | 197 | 198 | 201 | 200 | 198 | 199 | 203
  5-9Y, 207082_KE_Kombewa | 96 | 81 | 94 | 79 | 78 | 74 | 58 | 55 | 60 | 67
  5-9Y, 207083_GH_Kintampo: number analyzed (Participants) | 200 | 200 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  5-9Y, 207083_GH_Kintampo | 115 | 103 |  |  |  |  |  |  |  |
  5-9Y, 207083_GH_Kintampo_EXP: number analyzed (Participants) | 0 | 0 | 199 | 202 | 200 | 198 | 200 | 202 | 200 | 200
  5-9Y, 207083_GH_Kintampo_EXP |  |  | 108 | 83 | 73 | 66 | 58 | 49 | 39 | 29
  5-9Y, 207083_GH_Kintampo_UNEXP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 199 | 201 | 197 | 201 | 201
  5-9Y, 207083_GH_Kintampo_UNEXP |  |  |  |  |  | 74 | 67 | 41 | 49 | 34
  5-9Y, 207084_SN_Keur Soce: number analyzed (Participants) | 200 | 203 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  5-9Y, 207084_SN_Keur Soce | 1 | 2 |  |  |  |  |  |  |  |
  5-9Y, 228607_GH_Navrongo_EXP: number analyzed (Participants) | 0 | 0 | 0 | 197 | 204 | 199 | 202 | 200 | 200 | 200
  5-9Y, 228607_GH_Navrongo_EXP |  |  |  | 69 | 70 | 65 | 58 | 55 | 49 | 52
  5-9Y, 228607_GH_Navrongo_UNEXP: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 200 | 199 | 201 | 201 | 193
  5-9Y, 228607_GH_Navrongo_UNEXP | 0 | 0 | 0 | 0 | 0 | 80 | 67 | 48 | 61 | 59
  5-9Y, 233149_MA_Mangochi: number analyzed (Participants) | 0 | 0 | 0 | 0 | 198 | 204 | 197 | 211 | 202 | 201
  5-9Y, 233149_MA_Mangochi |  |  |  |  | 47 | 47 | 24 | 44 | 51 | 36
  5-9Y, 233149_MA_Monkey Bay: number analyzed (Participants) | 0 | 0 | 0 | 0 | 203 | 200 | 201 | 194 | 202 | 196
  5-9Y, 233149_MA_Monkey Bay |  |  |  |  | 36 | 27 | 16 | 23 | 51 | 26
  5-9Y, 233150_MA_Chikwawa: number analyzed (Participants) | 0 | 0 | 0 | 0 | 192 | 0 | 206 | 202 | 201 | 200
  5-9Y, 233150_MA_Chikwawa |  |  |  |  | 36 | 0 | 54 | 22 | 10 | 13
  5-9Y, 233150_MA_St Monfort: number analyzed (Participants) | 0 | 0 | 0 | 0 | 195 | 0 | 199 | 198 | 201 | 202
  5-9Y, 233150_MA_St Monfort |  |  |  |  | 21 | 0 | 26 | 9 | 10 | 2
  5-9Y, 235578_KE_Bondo: number analyzed (Participants) | 0 | 0 | 0 | 0 | 206 | 208 | 199 | 201 | 200 | 200
  5-9Y, 235578_KE_Bondo |  |  |  |  | 64 | 80 | 65 | 64 | 50 | 42
  5-9Y, 235578_KE_Gem: number analyzed (Participants) | 0 | 0 | 0 | 0 | 197 | 195 | 202 | 201 | 202 | 200
  5-9Y, 235578_KE_Gem |  |  |  |  | 66 | 67 | 67 | 51 | 62 | 45
  5-9Y, 235579_KE_Nyando: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 203 | 205 | 194 | 197 | 192
  5-9Y, 235579_KE_Nyando |  |  |  |  |  | 70 | 59 | 33 | 51 | 50

14. Primary Outcome: Number of Participants Using Malaria Control Interventions: Bednet Usage and Type of Bednet
Description: The number of participants using malaria control interventions was summarized by: participants sleeping under a mosquito net the night before their visit, participants who have a new bednet (less than 1 year), participants who have a impregnated bednet (dipped in liquid to repel mosquitos after purchase), participants who have a pierced/torn bednet, participants with bednets classified by hole size (defined as holes big enough to let one finger go through) and number of holes (less than [<] 5 holes, more or equal [>=] to 5 holes, not applicable [NA] which is a participant who did not sleep under a bed net, missing confirmed [MC] which is a participant who slept under a mosquito net but who didn't answer to the question on holes).
Time Frame: At Day 1 (survey completion visit)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group
Number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
Participants
  Participant sleep under a mosquito net night before visit | 3768 | 3628 | 2152 | 2733 | 4805 | 5140 | 6281 | 6312 | 6125 | 6161
  New bednet [less than 1 year] | 2524 | 2081 | 1552 | 1843 | 2897 | 2292 | 3829 | 4086 | 2986 | 3889
  Impregnated [dipped in liquid to repel mosquitos after purchase] Bednet | 2590 | 2825 | 1359 | 2457 | 4201 | 4458 | 5623 | 5343 | 5397 | 5449
  Pierced/torn Bednet | 906 | 872 | 431 | 500 | 1805 | 2142 | 1874 | 2017 | 2487 | 1761
  How many holes of size, Less than 5 | 435 | 347 | 261 | 398 | 1271 | 1427 | 1255 | 1455 | 1791 | 1189
  How many holes of size, More or equal to 5 | 471 | 525 | 170 | 102 | 534 | 715 | 619 | 562 | 696 | 572
  How many holes of size, NA | 3302 | 3327 | 1968 | 2500 | 3572 | 3845 | 5366 | 5200 | 4716 | 5441
  How many holes of size, MC: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 7241 | 0 | 0 | 0
  How many holes of size, MC |  |  |  |  |  |  | 1 |  |  |

15. Primary Outcome: Number of Participants Using Malaria Control Interventions: Mosquito Coils, Insecticide Sprays, Commercial Repellants, Traditional Repellants and Indoor Residual Sprays
Description: The number of participants using malaria control interventions was summarized by: mosquito coils, insecticide sprays, commercial repellants, traditional repellants and indoor residual sprays (in the past 12 months, 1 to 12 months, NA [the participant didn't use the residual spray], missing [participant used spray but didn't answer to how long ago]).
Time Frame: At Day 1 (survey completion visit)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group
Number analyzed (Participants) | 4208 | 4199 | 2399 | 3000 | 5377 | 5987 | 7241 | 7217 | 7203 | 7202
Participants
  Use of Mosquito coils | 246 | 305 | 150 | 359 | 452 | 808 | 1137 | 1205 | 1379 | 1514
  Use of Insecticide sprays | 52 | 65 | 44 | 118 | 119 | 230 | 265 | 325 | 253 | 247
  Use of Commercial Repellents | 56 | 22 | 14 | 19 | 22 | 50 | 68 | 114 | 103 | 60
  Use of Traditional Repellents | 122 | 106 | 1 | 8 | 103 | 28 | 134 | 74 | 149 | 108
  Use of indoor residual spray (IRS) in past 12 months | 300 | 42 | 5 | 279 | 293 | 1749 | 1797 | 1819 | 1978 | 1932
  Use of IRS 1 month ago | 1 | 15 | 1 | 208 | 17 | 21 | 1 | 18 | 35 | 8
  Use of IRS 2 month ago | 161 | 7 | 2 | 38 | 20 | 14 | 5 | 7 | 51 | 17
  Use of IRS 3 month ago | 124 | 8 | 0 | 13 | 35 | 45 | 45 | 52 | 155 | 98
  Use of IRS 4 month ago | 1 | 1 | 0 | 1 | 58 | 134 | 102 | 59 | 248 | 179
  Use of IRS 5 month ago | 0 | 0 | 1 | 4 | 69 | 274 | 420 | 187 | 338 | 222
  Use of IRS 6 month ago | 2 | 0 | 0 | 4 | 44 | 452 | 665 | 557 | 434 | 148
  Use of IRS 7 month ago | 0 | 0 | 0 | 0 | 17 | 359 | 519 | 555 | 443 | 407
  Use of IRS 8 month ago | 1 | 1 | 0 | 0 | 13 | 330 | 33 | 309 | 187 | 773
  Use of IRS 9 month ago | 10 | 5 | 1 | 0 | 7 | 114 | 1 | 64 | 75 | 75
  Use of IRS 10 month ago | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 10 | 0
  Use of IRS 11 month ago | 0 | 3 | 0 | 0 | 3 | 3 | 0 | 7 | 1 | 5
  Use of IRS 12 month ago | 0 | 2 | 0 | 11 | 5 | 2 | 5 | 3 | 1 | 0
  Use of IRS, NA | 3908 | 4175 | 2394 | 2721 | 5084 | 4238 | 5444 | 5398 | 5221 | 5270
  Missing: number analyzed (Participants) | 0 | 0 | 0 | 0 | 5377 | 0 | 0 | 0 | 7203 | 0
  Missing |  |  |  |  | 2 |  |  |  | 4 |

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and all-cause mortality were collected from Year 1 to Year 10
Description: According to the pre-specified protocol, only serious adverse events were collected. Since no other adverse events were captured in this study, the total number of participants at risk or affected by non-serious adverse events is zero. The analysis was performed on the Total Effective Cohort.
Arm/Group | Survey 1 Group | Survey 2 Group | Survey 3 Group | Survey 4 Group | Survey 5 Group | Survey 6 Group | Survey 7 Group | Survey 8 Group | Survey 9 Group | Survey 10 Group
All-Cause Mortality (participants affected / at risk) | 0/4214 | 0/4204 | 0/2400 | 0/3003 | 0/5417 | 0/5991 | 0/7246 | 0/7220 | 0/7203 | 0/7202
Serious Adverse Events (participants affected / at risk) | 0/4214 | 0/4204 | 0/2400 | 0/3003 | 0/5417 | 0/5991 | 0/7246 | 0/7220 | 0/7203 | 0/7202
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/04/NCT02251704/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/04/NCT02251704/SAP_001.pdf